| Division | : Worldwide Development |
|------------------|-------------------------------|
| Information Type | : Reporting and Analysis Plan |

Title : Reporting and Analysis Plan for Study 201881: A
Randomized, Double-blind, Sponsor un-Blinded, Placebocontrolled, Phase 2a Crossover Study to Evaluate the Effect
of the TRPV4 Channel Blocker, GSK2798745, on Pulmonary
Gas Transfer and Respiration in Patients with Congestive
Heart Failure

Compound Number : GSK2798745

Effective Date : 18-OCT-2017

### **Description:**

- The purpose of this reporting and analysis plan (RAP) is to describe the final planned analyses and output to be included in the Clinical Study Report for Study 201881.
- This RAP is intended to describe the planned efficacy, safety & tolerability, pharmacokinetics analysis required for the study.
- This document will be provided to the study team members to convey the content of the final Statistical Analysis Complete (SAC) Deliverable.

### Author's Name and Functional Area:

| PPD | 18-OCT-2017 |
|----------------------------------------------|-------------|
| Principal Statistician (Clinical Statistics) | 18-OC1-2017 |
| PPD | 18-OCT-2017 |
| Statistician (Clinical Statistics) | 16-001-2017 |
| PPD | 19 OCT 2017 |
| Director, (CPMS) | 18-OCT-2017 |

### Approved by:

| PPD | 19 OCT 2017 |
|-----------------------------------|-------------|
| TA Director (Clinical Statistics) | 18-OCT-2017 |

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | REPO | RTING & A | NALYSIS PLAN SYNPOSIS | 4 |
| 2. | RAP A | MENDME | NTS | 4 |
| 3. | SUMM | ARY OF K | EY PROTOCOL INFORMATION | 5 |
| • | 3.1. | | to the Protocol Defined Statistical Analysis Plan | |
| | 3.2. | | ective(s) and Endpoint(s) | |
| | 3.3. | | sign | |
| | 3.4. | Statistical | Hypotheses | 7 |
| 4. | PLAN | NED ANAL | YSES | <mark>7</mark> |
| | 4.1. | | nalyses | |
| | 4.2. | Final Anal | yses | 8 |
| 5. | ANALY | | JLATIONS | |
| | 5.1. | Protocol D | Deviations | 9 |
| 6. | _ | | SIDERATIONS FOR DATA ANALYSES AND DATA VENTIONS | 9 |
| 7. | | | TION ANALYSES | |
| | 7.1. | Planned A | Analyses Overview | 10 |
| 8. | PRIMA | RY STATI | STICAL ANALYSES | 11 |
| | 8.1. | | nalyses | |
| | | 8.1.1. | Overview of Planned Efficacy Analyses | 11 |
| | | 8.1.2. | Statistical Model | 12 |
| 9. | SECO | NDARY ST | TATISTICAL ANALYSES | 12 |
| | 9.1. | | nalyses | |
| | | | Overview of Planned Efficacy Analyses | |
| | 9.2. | | alyses | |
| | 9.3. | | Overview of Planned Analyses | |
| | 9.3. | 9.3.1. ( | okinetic Analyses Overview of Planned Pharmacokinetic Analyses | 15 |
| | | | Drug Concentration Measures | |
| | | | Pharmacokinetic Parameters | |
| | | ( | 9.3.3.1. Deriving Pharmacokinetic Parameters | 16 |
| 10. | REFE | RENCES | | 18 |
| 11 | A DDEN | IDICES | | 10 |
| 11. | 11.1. | | 1: Protocol Deviation Definitions for Per Protocol | 19 |
| | | Population | າ | |
| | | 11.1.1. | Exclusions from Per Protocol Population | 20 |
| | 11.2. | | 2: Time and Events | |
| | Appen 11.3. | | and Events | |
| | 11.3. | | Treatment Phases | |

### **CONFIDENTIAL**

| | 11.3.2. | Treatment States | |
|---|---|---|---|
| | 11.3.3. | Treatment States for AE Data | 25 |
| 11.4. | Appendix | x 4: Data Display Standards & Handling Conventions | 26 |
| | 11.4.1. | Study Treatment & Sub-group Display Descriptors | |
| | 11.4.2. | Baseline Definition & Derivations | |
| | | 11.4.2.1. Baseline Definitions | 26 |
| | | 11.4.2.2. Derivations and Handling of Missing Baseline | |
| | | Data | 26 |
| | 11.4.3. | Reporting Process & Standards | 26 |
| 11.5. | Appendix | x 5: Derived and Transformed Data | |
| | 11.5.1. | General | |
| | 11.5.2. | Study Population | 29 |
| | 11.5.3. | Safety | |
| 11.6. | Appendix | x 6: Premature Withdrawals & Handling of Missing Data | 31 |
| | 11.6.1. | Premature Withdrawals | |
| | 11.6.2. | Handling of Missing Data | |
| | | 11.6.2.1. Handling of Missing Dates | |
| | | 11.6.2.2. Handling of Partial Dates | |
| 11.7. | Appendix | x 7: Values of Potential Clinical Importance | |
| | | Laboratory Values | |
| | 11.7.2. | • | |
| | 11.7.3. | Vital Signs | 34 |
| 11.8. | Appendix | x 8: Laboratory A&R Dataset Details | |
| 11.9. | | x 9: Biomarker A&R Dataset Details | |
| 11.10. | | x 10 – Abbreviations & Trade Marks | |
| | | Abbreviations | |
| | | Trademarks | |
| 11.13. | | x 11: List of Data Displays | |
| | | Data Display Numbering | |
| | | Deliverable [Priority] | |
| | | Mock Example Numbering | |
| | | Study Population Tables | |
| | | Efficacy Tables | |
| | | Efficacy Figures | |
| | | Safety Tables | |
| | | Pharmacokinetic Tables | |
| | | Pharmacokinetic Figures | |
| | | OICH Listings | |
| | | .Non-ICH Listings | |
| 11 14 | | x 12: Example Mock Shells for Data Displays | |

## 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | This RAP details all planned analyses and outputs required for the final Clinical Study Report (CSR) of Study 201881. |
| Protocol | This RAP is based on the protocol amendment 02 (Dated: 19-APR-2016) for Study 201881 [GlaxoSmithKline Document Number: ]. |
| Primary<br>Objective | To assess the effect of GSK2798745 on pulmonary gas transfer |
| Primary<br>Endpoint | Change in the diffusing capacity for carbon monoxide (DLco) |
| Study<br>Design | This is a randomized, double-blind, sponsor-unblinded, placebo-controlled, 2X2 crossover study in adults with heart failure. |
| | 12 subjects are planned to complete both treatment periods. Additional subjects up to 24 in total maybe needed based on interim decision |
| Planned | Interim analyses are detailed within Section 4.1 where applicable. |
| Analyses | All decisions regarding final analysis, as defined in this RAP document, will be made prior to Database Freeze (unblinding) of the study data. |
| Primary<br>Analysis<br>Population | <ul> <li>The 'All Subjects' Population is defined as all randomized subjects who receive at least one dose of study medication.</li> <li>The 'Analysis Population' is defined as subjects in the 'All Subjects' population having baseline and post-baseline assessments of the endpoint of interest for both periods.</li> <li>The 'Per Protocol' Population will consist of any 'Analysis Population' subjects who are compliant with protocol-specific criteria. Subjects with specified protocol deviations will be excluded.</li> <li>The 'Pharmacokinetic (PK)' Population is defined as subjects for whom a pharmacokinetic sample was obtained and analysed.</li> </ul> |
| Hypothesis | <ul> <li>An estimation approach will be used for the comparison between GSK2798745 treatment<br/>and placebo for the change from baseline in DLco at Day 4 and Day 7. Point estimates<br/>and associated 95% confidence intervals for the differences in means will be constructed<br/>to provide a plausible range of values for the true comparisons of interest.</li> </ul> |
| Primary<br>Analyses | • Profiles for DLco will be summarized and presented graphically by treatment group and visits as appropriate for the data. The change from baseline in DLco at Day 4, Day 6 and Day 7 will be calculated and summarized in tabular format and/or graphically by treatment. For the change from baseline in DLco, a statistical analysis will be performed using a mixed effect model with repeated measures with a fixed effect term for treatment, period and day, with a random effect for subject, and baseline as a covariate, if data permit. Point estimates and associated 95% confidence intervals will be constructed for the differences between the active treatment and placebo. |

## 2. RAP AMENDMENTS

18- Oct-2017: Given the decision to not continue the TRPV4 HF work on this asset, the exploratory Bayesian analysis was removed. Addition of some FDAAA required tables, listing, and figures.

## 3. SUMMARY OF KEY PROTOCOL INFORMATION

## 3.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol amendment 02 (Dated: 19-APR-2016).

## 3.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To assess the effect of<br>GSK2798745 on pulmonary gas<br>transfer | Change in the diffusing capacity for carbon monoxide (DLco) |
| Secondary Objectives | Secondary Endpoints |
| To assess the effect of<br>GSK2798745 on alveolar-capillary<br>conductance (DM) | Change in the diffusing capacity for nitric oxide (DLno), membrane conductance (DM), and capillary blood volume (Vc) |
| To assess the effect of<br>GSK2798745 on pulmonary gas<br>transfer following exercise and<br>following an intravenous saline<br>infusion | Change in diffusing capacity for carbon monoxide (DLco) |
| To evaluate the effect of<br>GSK2798745 on ventilatory<br>efficiency | Change in the VE/VCO2 slope determined during a standardized 3-minute step test |
| To evaluate the effect of<br>GSK2798745 on pulmonary<br>function | Changes in spirometry measures including forced vital capacity (FVC) and forced expiratory volume in 1 second (FEV1) as well as forced expiratory flows, FEF25-75 FEF50, and FEF75 |
| | <ul> <li>Change in functional residual capacity (FRC) and<br/>end-expiratory lung volume (EELV) measured by<br/>body plethysmograph</li> </ul> |
| To assess the effect of<br>GSK2798745 on dyspnea | Change in dyspnea score |
| To assess the effect of<br>GSK2798745 on respiratory rate | Change in respiratory rate continuously measured by body sensor (Preventice Body Guardian) |
| To evaluate the safety and tolerability of repeat administration of GSK2798745 | Clinical monitoring of vital signs, ECGs, and clinical laboratory safety data, including LFTs and troponin as well as reporting of adverse events (AEs) |
| To assess the effect of<br>GSK2798745 on quality of life | Change in SF-36 acute score |
| To characterize the pharmacokinetic profile of GSK2798745 in subjects with heart failure | <ul> <li>Area under the concentration time curve (AUC),<br/>maximum drug concentration (Cmax), time to<br/>maximum observed plasma concentration (tmax),<br/>and elimination halflife (T½)</li> </ul> |

| Objectives | Endpoints |
|---|---|
| Exploratory Objectives | Exploratory Endpoints |
| To determine the effect of<br>GSK2798745 on oxygen saturation | Change in minimum O2 saturation measured during polysomnography |
| To assess effect of GSK2798745<br>on sleep disordered breathing<br>patterns | <ul> <li>Change in apnea-hypopnea index (AHI) determined by polysomnography</li> <li>Change in the central, obstructive and mixed apnea indexes as determined by polysomnography</li> <li>Change in respiratory temporal dynamics during inhouse sleep apnea evaluation</li> </ul> |
| To determine whether GSK2798745 affects sleep- disordered breathing leading to an improvement in sympathoadrenal activity | Change in plasma and urinary catecholamine concentrations in subjects with sleep-disordered breathing |
| To determine whether GSK2798745 affects electrocardiographic parameters | Changes in time and frequency domain analyses of<br>ECG: HR variability to define sympathetic activity |
| To explore the impact of<br>GSK2798745 on the exposure of<br>HMG-CoA reductase inhibitors | AUC of HMG-CoA reductase inhibitors and their key metabolites |

## 3.3. Study Design



| Overview of Study Design and Key Features | |
|---|---|
| · | <ul> <li>study will be conducted at multiple centers.</li> <li>Subjects have an at least 3 month history of HF, be a NYHA Class II-IV,a NT-proBNP of greater than 400 pg/ml within the last 6 months and a % predicted DLco of &lt; 80% at screening.</li> </ul> |
| Dosing | <ul> <li>Subjects are dosed once daily for 7 days. Then there is a wash out<br/>period of at least 14 days, followed by another 7 days of once daily<br/>dosing.</li> </ul> |
| Treatment<br>Assignment | <ul> <li>Eligible subjects will be randomized to one of two treatment sequences.</li> <li>A sufficient number of subjects with heart failure will be enrolled so that 12 subjects complete the two study periods and critical assessments.</li> <li>Subjects will receive either GSK2798745 or placebo once daily for a period of 7 days.</li> <li>After at least a 14-day washout period (preferably not greater than 30 days from last dose in Period I), subjects will participate in a second, identical 7-day study period and receive the alternate study medication.</li> </ul> |
| Interim Analysis | <ul> <li>After approximately 5-6 subjects complete both study periods, a sponsor unblinded interim analysis will be performed.</li> <li>After approximately 9 subjects complete both study periods, a sponsor unblinded interim analysis will be performed.</li> <li>After 12 subjects complete both study periods, prior to SAC, an interim analysis will be performed to determine if additional subjects will be enrolled in the study (up to 24 subjects). Full details are in Section 3.1</li> </ul> |

## 3.4. Statistical Hypotheses

An estimation approach will be used for the comparison between GSK2798745 treatment and placebo for the change from baseline in DLCo at day 4 and day 7. Point estimates and associated 95% confidence intervals for the differences in means will be constructed to provide a plausible range of values for the true comparisons of interest.

### 4. PLANNED ANALYSES

## 4.1. Interim Analyses

- There will be ongoing data reviews by the study team of the un-blinded safety and pharmacokinetics data throughout the trial progression.
- After approximately 6 Subjects complete both study periods, a sponsor un-blinded interim analysis will be performed on DLco and other variables of potential clinical relevance. The programming code for this interim analysis will be provided by the study statistician.

- After approximately 9 subject complete both study periods, a sponsor un-blinded interim analysis will be performed.
- After 12 subjects complete both study periods, prior to DBF, a sponsor un-blinded interim analysis will be performed on DLco.

A Bayesian predictive probability of change in DLco with 18 patients will be calculated, and the intra-subject variability will be estimated. These analyses will inform a decision to enrol up to 12 additional subjects.

Given the decision to not continue the TRPV4 HF work on this asset, the Bayesian prediction was performed on 10 subjects and a decision was made to only enrol one more patient. Therefore, an interim analysis will not be performed on 12 subjects.

### 4.2. Final Analyses

The final planned analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol.
- 2. All required database cleaning activities have completed the final database release and database freeze has been declared by Data Management.
- 3. All criteria for unblinding the randomisation codes have been met.
- 4. Randomisation codes have been distributed accordingly to RandAll NG procedures.

## 5. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All<br>Subjects | <ul> <li>The 'All Subjects' Population is defined as all<br/>randomized subjects who receive at least one dose of<br/>study medication.</li> </ul> | <ul><li>Study Population</li><li>Safety/tolerability</li></ul> |
| Enrolled | All participants who sign informed consent and for whom a record exists on the study database. This population will be used for the tables/listings of reasons for withdrawal before randomization and listings of AEs and SAEs for non-randomized participants. | <ul> <li>Subject Disposition</li> <li>Reasons for<br/>withdrawal before<br/>randomization.</li> </ul> |
| | | <ul> <li>Inclusion, exclusion,<br/>and randomization<br/>criteria deviations</li> </ul> |
| Analysis<br>Population | <ul> <li>Subjects in the 'All Subjects' population having baseline<br/>and post-baseline assessments of the endpoint of interest<br/>for both periods</li> </ul> | <ul><li>Efficacy</li><li>PD/Biomarker</li></ul> |
| Screening Population | <ul> <li>The "Screening Population" is defined as all subjects who<br/>were screened as potential patients for the trial</li> </ul> | Screen Failure |
| Per<br>Protocol | <ul> <li>Any 'Analysis Population' subjects who are compliant<br/>with protocol-specific criteria. Subjects with specified<br/>protocol deviations will be excluded.</li> </ul> | Efficacy |
| PK<br>Population | • This population will include all subjects in the Safety Population for whom a pharmacokinetic blood sample was obtained and assayed. | • Concentration data summaries, |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| | | listings, and<br>graphs (including<br>concentration-time<br>profiles as<br>appropriate) |
| PK<br>Parameter<br>Population | This population will include all subjects in the PK Concentration Population for whom valid and evaluable pharmacokinetic parameters were derived. | • Listings, summary and analyses of PK parameters |

#### NOTE:

 Please refer to Section 11.13 Appendix 11: List of Data Displays which details the population to be used for each display being generated.

### 5.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.
- Important deviations which result in exclusion from the analysis population will also be summarised and listed. (Please refer to Appendix 1: Protocol Deviation Definitions for Per Protocol Population).
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.

# 6. GENERAL CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

- There are no planned examinations of covariates. The only subgroups analysis planned is by site.
- There are no planned adjustments for multiple comparisons or multiplicity.

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| 11.1 | Appendix 1: Protocol Deviation Definitions for Per Protocol Population |
| 11.2 | Appendix 2: Time and Events |

| Section | Component |
|---------|--------------------------------------------------------------|
| 11.3 | Appendix 3: Treatment States and Phases |
| 11.4 | Appendix 4: Data Display Standards & Handling Conventions |
| 11.5 | Appendix 5: Derived and Transformed Data |
| 11.6 | Appendix 6: Premature Withdrawals & Handling of Missing Data |
| 11.7 | Appendix 7: Values of Potential Clinical Importance |
| 11.8 | Appendix 8: Laboratory A&R (QUEST: LAB) Dataset Details |
| 11.9 | Appendix 9: Biomarker A&R Dataset Details |

## 7. STUDY POPULATION ANALYSES

## 7.1. Planned Analyses Overview

The study population analyses will be based on the "All Subjects" population, unless otherwise specified.

Table 2 provides an overview of the planned study population analyses with full details of data displays being presented in Appendix 11: List of Data Displays.

Table 2 Overview of Planned Study Population Analyses

| Display Type | Data l | Display's Gen | erated |
|---|---|---|---|
| | Figure | Table | Listing |
| Randomisation | | | |
| Randomisation | | | Υ |
| Subject Disposition | | | |
| Subject Disposition | | Υ | |
| Reasons for Screening Failures | | | Y |
| Reasons for Withdrawals | | Υ | Y |
| Important Protocol Deviations | | Υ | Y |
| Deviations Leading to Exclusions from PP Population | | Υ | Y |
| Inclusion and Exclusion Criteria Deviations | | | Υ |
| Demography | | | |
| Demographics Characteristics | | Υ | Υ |
| Race & Racial Combinations | | Υ | Υ |
| Study Populations | | Υ | |
| Medical Condition & Concomitant Medications | | | |
| Medical Conditions (Current/Past) | | Υ | Y |
| Concomitant Medication | | Y | Υ |

### 8. PRIMARY STATISTICAL ANALYSES

## 8.1. Efficacy Analyses

### 8.1.1. Overview of Planned Efficacy Analyses

The efficacy analyses will be based on the "Analysis Population", unless otherwise specified.

Table 3 provides an overview of the planned efficacy analyses with full details of data displays being presented in Appendix 11: List of Data Displays.

Table 3 Overview of Planned Efficacy Analyses

| ENDPOINT | Ab | solu | te | | Change from Baseline | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats | | Summary | | Individual | | Stats | | | Summary | | Indiv | idual | |
| | An | Analysis | | | | | | | Analysis | | | | | |
| | Т | F | L | T | F | F | Ш | Т | H | L | T | F | F | L |
| DLco | DLco | | | | | | | | | | | | | |
| Diffusing capacity for carbon monoxide (DLco) | Υ | | | Υ | Υ | | Υ | Υ | | | Υ | Υ | | Υ |

### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

### 8.1.2. Statistical Model

Analysis of variance (ANOVA) with repeated measure will be performed on DLco. The primary interested outcome is to compare the treatment effects of the two treatments, where the treatment effect is defined as the change of DLco at the end of each treatment period from the corresponding baseline. Methodological differences in how DLco is collected at the two site causes variance differences by site so it will not be possible to pool DLco values across sites.

The model assumes no cross-over effect. This assumption will be tested by the following code:

```
data results;
        set results;
        contrast = 0.5*(baseline_period1 - baseline_period2);
run;

proc ttest alpha=0.10;
    class seq;
    var contrast;
run;
```

Due to the small sample size, this test has a low power to detect cross-over effects, so the assumption will also be tested graphically by looking at a plot of measures overtime. If there are any departures from the distributional assumptions, alternative models will be explored using appropriately transformed data.

### 9. SECONDARY STATISTICAL ANALYSES

### 9.1. Efficacy Analyses

### 9.1.1. Overview of Planned Efficacy Analyses

The secondary efficacy analyses will be based on the "Analysis Population", unless otherwise specified.

The study is being conducted at two sites. One of these two sites does not have the ability to collect DLno, DM, and Vc. Summaries of DLno, DM, and Vc will only be performed for subjects at the site which this data is collected.

When calculating summary statistics for efficacy data, pooled summaries and summaries for each site individually will be generated. Patient ID's in the PPD are from the Mayo Clinic and patients ID's in the PPD are from Hennepin.

Table 4 provides an overview of the planned efficacy analyses with further details of data displays being presented in Appendix 11: List of Data Displays.

All change from baseline table, listing, and figures, use the baseline measured just prior to the period, (i.e. period 1 measurements use the baseline measured just prior to period 1 and period 2 measures use the baseline measured just prior to period 2), unless otherwise specified.

Statistical analysis (adjusted means and/or posterior means) will be performed on secondary endpoints as shown in Table 4

Table 4 Overview of Planned Efficacy Analyses

| Endpoint | | | Abs | olute | | | Change from Baseline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | ats<br>lysis | Sum | mary | Indiv | ridual | | ats<br>lysis | Sum | mary | Indiv | idual |
| | Т | F | T | F | F | L | Т | F | T | F | F | L |
| Diffusing capacity | Υ | | Υ | Υ | Υ | Υ | | | Υ | Υ | Υ | Υ |
| for nitric oxide | | | | | | | | | | | | |
| (DLno) | | | | | | | | | | | | |
| Membrane | Υ | | Υ | Υ | Υ | Υ | | | Υ | Υ | Υ | Υ |
| conductance (DM) | | | | | | | | | | | | |
| Capillary blood | Υ | | Υ | Υ | Υ | Υ | | | Υ | Υ | Υ | Υ |
| volume (Vc) | | | | | | | | | | | | |
| Dm/Vc | Υ | | Υ | | Υ | | | | Υ | | | |
| Diffusing capacity | | | Υ | Υ | Υ | Υ | | | Υ | Υ | Υ | Υ |
| for carbon | | | | | | | | | | | | |
| monoxide (DLco) | | | | | | | | | | | | |
| following exercise | | | | | | | | | | | | |
| Diffusing capacity | | | Υ | Υ | Υ | Υ | | | Υ | Υ | Y* | Υ |
| for carbon | | | | | | | | | | | | |
| monoxide (DLco) | | | | | | | | | | | | |
| following saline | | | | | | | | | | | | |
| infusion | | | | | | | | | | | | |
| VE/VCO <sub>2</sub> ratio | | | Υ | Υ | Υ | Υ | | | Υ | Υ | Υ | Υ |
| Forced vital | | | Υ | Υ | Υ | Υ | | | Υ | Υ | | Υ |
| capacity (FVC) | | | | | | | | | | | | |
| Forced expiratory | | | Υ | Υ | Υ | Υ | | | Υ | Υ | | Υ |
| volume in 1 | | | | | | | | | | | | |
| second (FEV1) | | | | | | | | | | | | |
| Forced expiratory | | | Υ | Υ | Υ | Υ | | | Υ | Υ | | Υ |
| flow, FEF25-75 | | | | | | | | | | | | |
| Forced expiratory | | | Υ | Υ | Υ | Υ | | | Υ | Υ | | Υ |
| flow, FEF50 | | | | | | | | | | | | |
| Forced expiratory | | | Υ | Υ | Υ | Υ | | | Υ | Υ | | Υ |
| flow, FEF75 | | | | \ , . | | | | | | | | |
| Respiratory rate | | | Υ | Υ | Υ | | | | | | | |
| (Preventice Body | | | | | | | | | | | | |
| Guardian) | | | | | | | | | | | | |
| Troponin | | | Υ | | | Y | | | Υ | | | Υ |
| SF-36 acute score | | | Υ | | | Υ | | | Υ | Υ | | |
| Dyspnea score | | | Υ | | | Υ | | | Υ | Υ | | Υ |

<sup>\*</sup>Change from value is calculated by taking the post-saline measure to the prior saline measure

## 9.2. Safety Analyses

## 9.2.1. Overview of Planned Analyses

The safety analyses will be based on the "All Subjects" population, unless otherwise specified.

Table 5 provides an overview of the planned analyses with further details of data displays being presented in Appendix 11: List of Data Displays.

Table 5 Overview of Planned Safety Analyses

| Endpoint | | P | bsolute | | ( | Change fro | m Baselin | е |
|---|---|---|---|---|---|---|---|---|
| | Sum | mary | In | dividual | Sum | mary | Indiv | idual |
| | T | F | F | L | Т | F | F | L |
| Exposure | | | | | | | | |
| Extent of Exposure | Υ | | | Υ | | | | |
| Adverse Events | | | | | | | | |
| All AE's [1] | Υ | | | Υ | | | | |
| Common AE's | Υ | | | | | | | |
| All Drug-Related AE's | Υ | | | Υ | | | | |
| Serious AE's | Υ | | | Y | | | | |
| Withdrawal AE's | Υ | | | Y | | | | |
| C-SSR | | | | Y | | | | |
| SNAQ | | | | Y | | | | |
| Audiometry | | | | Y | | | | |
| Laboratory Values | | | | | | | | |
| Clinical Chemistry [2] [3] | Υ | | | Υ | Υ | | | Υ |
| LFT's | Υ | | | Υ | | | | |
| Hematology /Coagulation [2] [3] | | | | Υ | Y | | | Υ |
| ECG's | | | | | | | | |
| ECG Findings | Υ | | | Υ | | | | |
| ECG Values | | | | | Y | | | |
| Vital Signs | | | | | | | | |
| Vitals Values | Υ | | | Υ | Υ | | | Υ |

| Endpoint | | Α | bsolute | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| | Sum | mary | In | dividual | Sum | mary | Individual | |
| | T | F | F | L | Т | F | F | L |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- Listings will include subject's numbers for individual AE's & AE system organ classes, preferred terms and verbatim text.
- 2. Chemistry & haematology summaries will include both changes from baseline & results by PCI criteria.
- 3. Listings of chemistry and haematology data for subjects with abnormalities of PCI will be listed.
- 4. Urinalysis summaries will include changes from baseline results by dipstick categories.

### 9.3. Pharmacokinetic Analyses

### 9.3.1. Overview of Planned Pharmacokinetic Analyses

The pharmacokinetic (PK) analyses will be based on the "Pharmacokinetic Parameter" population, unless otherwise specified.

Table 6 provides an overview of the planned analyses with full details being presented in Appendix 11: List of Data Displays.

Table 6 Overview of Planned Pharmacokinetic Analyses

| Endpoints | | Untrans | formed | | Log-Transformed | | | |
|---|---|---|---|---|---|---|---|---|
| | Summary | | Indiv | idual | Summary | | Individual | |
| | F | T | F | L | F | Т | F | L |
| Plasma Drug Concentrations | <b>Y</b> [2][3] | Υ [3] | Υ[1] | Υ | <b>Y</b> [2][3] | | | |
| Derived PK Parameters | | Υ [3] | | Υ | | Y [3] | | |

### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. Linear and Semi-Log plots will be created on the same display.
- 2. Mean (Linear and Semi-Log on same display) and Median (Linear and Semi-Log on same display) plots will be created.
- 3. Displays generated using the 'PK parameter populations.

## 9.3.2. Drug Concentration Measures

Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 11.4.3 Reporting Process & Standards).

### 9.3.3. Pharmacokinetic Parameters

## 9.3.3.1. Deriving Pharmacokinetic Parameters

- Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 11.4.3 Reporting Process & Standards).
- The pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using Win Nonlin.
- All calculations of non-compartmental parameters will be based on actual sampling times.

## Table 7 Derived Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| First and Se | cond last Dose in each treatment period as data permit |
| AUC(0-tau) | Area under the concentration-time curve over the dosing interval after first and last dose |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data on Day 1 and Day 7. |
| tmax | Time to reach Cmax, determined directly from the concentration-time data. |
| If Assessab | le |
| Lamda_z | Terminal phase rate constant |
| t½ | Apparent terminal half-life will be calculated as: |
| | $t\frac{1}{2} = \ln 2 / \text{Lambda}_z$ |

## NOTES:

Additional parameters may be included as required.

## 10. REFERENCES

GlaxoSmithKline Document Number 2014N221874\_02: A Randomized, Double-blind, Sponsor unOblinded, Placebo-controlled, Phase 2a Crossover Study to Evaluate the Effect of the TRPV4 Channel Blocker, GSK2798745, on Pulmonary Gas Transfer and Respiration in Patients with Congestive Heart Failure. Effective date: 19-APR-2016

## 11. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 5 | : Analysis Populations |
| Section 11.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| RAP Section 6 | General Considerations for Data Analyses & Data Handling Conventions |
| Section 11.2 | Appendix 2: Time and Events |
| Section 11.3 | Appendix 3: Treatment States & Phases |
| Section 11.4 | <ul> <li>Appendix 4: Data Display Standards &amp; Handling Conventions</li> <li>Study Treatment &amp; Sub-group Display Descriptors</li> <li>Baseline Definitions &amp; Derivations</li> <li>Reporting Process &amp; Standards</li> </ul> |
| Section 11.5 | <ul> <li>Appendix 5: Derived and Transformed Data</li> <li>General, Study Population &amp; Safety</li> <li>Efficacy</li> <li>Pharmacokinetic</li> <li>Pharmacodynamic / Biomarkers</li> </ul> |
| Section 11.6 | Appendix 6: Premature Withdrawals & Handling of Missing Data • Handling of Missing Dates • Handling of Partial Dates |
| Section 11.7 | Appendix 7: Values of Potential Clinical Importance Laboratory Values ECG's Vital Signs |
| Section 11.8 | Appendix 8 : Laboratory A&R Datasets |
| Section 11.9 | Appendix 9 : Biomarker A&R Datasets |
| Other RAP App | endices |
| Section 11.10 | Appendix 10: Abbreviations & Trade Marks |
| Section 11.13 | Appendix 11: List of Data Displays |
| Section 0 | Appendix 12: Example Mock Shells for Data Displays |

# 11.1. Appendix 1: Protocol Deviation Definitions for Per Protocol Population

## 11.1.1. Exclusions from Per Protocol Population

A subject meeting any of the following criteria will be excluded from the Per Protocol population:

| Number | Exclusion Description |
|--------|--------------------------------------------------|
| 01 | Subject takes prohibited Concomitant Medications |
| 02 | Others as defined in the PDMP |

# 11.2. Appendix 2: Time and Events

# Appendix 2: Time and Events

| | Screening<br>Period | | | | Tre | atment Perio | ods I and II ( | Day) | | | | Follow-up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Day -25 to<br>Day -1 prior<br>to Period I | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 14 ± 4 days<br>after last<br>dose of<br>study<br>medication |
| Informed consent | X | | | | | | | | | | | |
| Inclusion and exclusion criteria | Х | | | | | | | | | | | |
| Demography | Х | | | | | | | | | | | |
| Full physical examination including height & weight | Х | | | | | | | | | | | |
| Brief physical exam including weight | | Х | | | | Х | | | Х | | | Х |
| Medical history/Medication history | Х | | | | | | | | | | | |
| Hepatitis B & C screen | Х | | | | | | | | | | | |
| Echocardiogram | X | | | | | | | | | | | |
| Urine drug and alcohol breath test | Х | Χ | | | | | | | | | | |
| Clinical lab<br>assessments <sup>14</sup> | Х | Х | | | | Х | | | Х | | | Х |
| NT-proBNP | Х | Χ | | | | | | | Χ | | | |
| Serum CTX <sup>11</sup> | | Χ | | | | | | | Х | | | |
| Fecal Occult Blood<br>Test <sup>12</sup> | Х | | | | | | | | Х | | | |
| Pharmacokinetic sample <sup>1</sup> | | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | Х | |
| Digoxin sample <sup>2</sup> | | Χ | Χ | Χ | Χ | Х | Χ | Χ | Х | | | Х |
| Troponin | X | Х | | Х | | Х | | | Х | | | Х |
| DLco/DLno <sup>10</sup> | Χ | Χ | | | | Х | Х | X | Х | | | Х |
| 12-lead ECG/<br>time & frequency<br>domains <sup>3</sup> | X <sub>9</sub> | X <sup>9</sup> | | | | х | | | Х | | | х |

| | Screening<br>Period | | | | Tre | eatment Peri | ods I and II ( | Day) | | | | Follow-up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Day -25 to<br>Day -1 prior<br>to Period I | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 14 ± 4 days<br>after last<br>dose of<br>study<br>medication |
| Vital signs | Х | Χ | Х | Х | Х | Х | Х | Х | Х | | | Х |
| Weight | | | Х | Х | Х | | Х | Х | | | | |
| Genetic sample | | | | For subject | ts who provid | de consent, s | ample collect | ed after start | of treatment | | • | |
| Study treatment <sup>4</sup> | | | Х | Χ | X | Χ | X | Х | Х | | | |
| AE/SAE review | | Χ | <b>←====</b> | ======= | | | | | <del>-</del> | | | Х |
| Concomitant med review | | Χ | <b>←====</b> | | | | | | <del>-</del> | | | Х |
| Pulmonary function tests | | Χ | | | | Х | | | Х | | | Х |
| Step exercise test/breath- | | Х | | | | | | | Х | | | Х |
| by-breath gas exchange | | | | | | | | | | | | |
| Dyspnea assessment | | Χ | | | | | Χ | | Х | | | X |
| Orthopnea | | | | | | | Χ | | | | | |
| SF-36 Acute | | Χ | | | | | | | Х | | | X |
| Polysomnography including oximetry (Sleep Apnea Clinic) <sup>5,13</sup> | | <b>←==</b> = | =====> | | | | | <b>←==</b> = | =====> | | | |
| Plasma and 8-hour urine catecholamines <sup>6</sup> | | Χ | | | | | | Х | | | | |
| Saline infusion | | | | | | | Χ | Χ | | | | |
| Admission to CRU <sup>7</sup> | | | Х | | | | | | | | | |
| Discharge from CRU <sup>7</sup> | | | | | Х | | | | | | | |
| Meals <sup>8</sup> | | Χ | Х | Х | Х | Х | Χ | Χ | Х | | | |
| Appetite Assessment (SNAQ) | | Х | | | | Х | | | Х | | | Х |
| CSSRS (Suicidality) | | Χ | | | | | | | Х | | | Х |
| Audiometry | | X <sup>13</sup> | | | | | | | Х | | | Х |
| BodyGuardian Monitor (Preventice) | | <b>←====</b> | ======= | ======= | ===Continuo | ous===== | ======= | ======= | <del>-</del> | | | |

- 1. Pharmacokinetic samples to determine GSK2798745 and any metabolite(s) concentrations will be obtained at the following times on Day 1 of each treatment period: Predose, 0.5, 1, 1.5, 2, 3, 5, 8 and 12 hours and at the following times on Day 7 of each treatment period: Predose, 0.5, 1, 1.5, 2, 3, and 5 and 10 hours. On Day 2 of each treatment period, samples will be collected predose and at 12 hours post dose. On Days 3 through 6, PK samples will be collected predose. On Days 8 and 9, samples will be collected at 24 and 48 hours, respectively, after the last dose of study medication administered on Day 7. The time points may be modified based on emerging data. Some of these timepoints may also be utilized to collect samples to determine concentrations of other medications (e.g., atorvastatin and/or simvastatin). See the SRM for detailed information.
- 2. Digoxin concentrations will be monitored only in those subjects who are taking digoxin
- 3. Time and frequency domains assessed by ECG obtained on Day -1 and Day 7
- 4. Subjects will remain in the CRU for a minimum of 4 hours after each administration of study medication. [Note: The first 6 subjects enrolled will remain in the CRU for 52 hours after the first dose of study medication in each period]
- 5. Only for subjects participating in the sub-study: At Day -1 of the first study period only, subjects will undergo an overnight sleep study. Only those subjects who are participating in the sub-study with sleep disordered breathing will undergo additional sleep studies on Day 6 of both study Periods I and II.
- 6. Only for subjects participating in the sub-study: Urinary norepinephrine (NE) and epinephrine (E) concentrations will be determined from 8-hour collections obtained during the overnight sleep study; urinary creatinine will also be measured to normalize the NE and E concentrations. A blood sample to determine plasma concentrations of NE and E will be obtained the morning after the sleep study between the hours of 9:00 am and 10:00 am after the subject has been supine for 20 minutes in a quiet room.
- 7. The first 6 subjects enrolled will remain in the CRU for two days (Day 1 and Day 2) after the first dose of study medication in each period.
- 8. Three meals per day will be provided by the dietary department either in the CRU or as a boxed meal(s) to take home.
- 9. ECGs to be performed in triplicate
- 10. On the days where exercise or the saline infusion is performed, DLco/DLno will be completed just prior to and after both exercise and the saline infusion.
- 11. Blood sample for analysis of Serum CTX must be collected when the subject is fasting.
- 12. Fecal Occult Blood Test (FOBT) cards will be provided to subjects at the end of the screening visit and must be completed and sent back to the laboratory prior to the baseline visit according to the laboratory's standard collection procedures. Similarly, subjects will be given FOBT cards at the end of the Day 7 visit of each study period with completion instructions.
- 13. Day -1 audiometry and sleep study assessments may be completed 7 days prior to Day -1.
- 14. Clinical laboratory assessments will be collected as a fasting sample.

## 11.3. Appendix 3: Treatment States and Phases

### 11.3.1. Treatment Phases

Assessments and events will be classified according to the time of occurrence relative to study treatment, unless otherwise specified.

| Treatment Phase | Definition |
|---|---|
| Pre-Treatment 1 | Date < Study Treatment Start Date for Period 1 |
| On-Treatment 1 | Study Treatment Start Date for Period 1≤ Date ≤ Study Treatment Stop Date for Period 1 |
| Post-Treatment 1 | Date > Study Treatment Stop Date for Period 1 |
| Pre-Treatment 2 | Date < Study Treatment Start Date for Period 2 |
| On-Treatment 2 | Study Treatment Start Date for Period 2 ≤ Date ≤ Study Treatment Stop Date for Period 2 |
| Post-Treatment 2 | Date > Study Treatment Stop Date for Period 2 |

### 11.3.2. Treatment States

Assessments and events will be classified according to time of occurrence relative to the start and/or stop date of the study treatment.

### 11.3.3. Treatment States for AE Data

| Treatment State | Definition |
|---|---|
| AE = Pre-Treatment | AE Start Date < Study Treatment Start Date |
| AE = On-Treatment | If AE onset date is on or after the treatment start date and on or before the treatment stop date. Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date [+ 1] |
| AE = Post-Treatment | If AE onset date is after the treatment stop date. AE Start Date > Study Treatment Stop Date + 1 |
| AE Onset Time<br>Since 1st Dose<br>(Days) | If Treatment Start Date > AE Onset Date : <b>= AE Onset Date - Treatment Start Date</b> If Treatment Start Date ≤ AE Onset Date : <b>= AE Onset Date - Treatment Start Date + 1</b> Missing otherwise |
| AE Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| AE = Drug-related | If relationship is marked 'YES' on [Inform/CRF OR value is missing. |

### NOTES:

• If the study treatment stop date is missing then the AE will be considered to be On-Treatment

# 11.4. Appendix 4: Data Display Standards & Handling Conventions

### 11.4.1. Study Treatment & Sub-group Display Descriptors

| Study Treatment Descriptions | | | |
|---|---|---|---|
| RandAll NG Data Displays for Reporting | | | |
| Code | Description | Description | Order |
| Α | GSK2798745 2.4 mg | GSK 2.4 mg | 2 |
| Р | Placebo | Placebo | 1 |

### 11.4.2. Baseline Definition & Derivations

### 11.4.2.1. Baseline Definitions

For all endpoints baseline value will be taken on Day -1 for each treatment period, unless otherwise specified.

### 11.4.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Dose Visit Value – The corresponding Baseline |
| [% Change from Baseline] | = [ (Post-Dose Visit Value – Baseline) / Baseline ] x 100] |

### NOTE:

- Unless otherwise specified, the baseline definitions specified in 11.4.2.1Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on all change from baseline displays.

### 11.4.3. Reporting Process & Standards

| Reporting Process | |
|---|---|
| Software | |
| The currently supported versions of Spotfire, SAS and R software will be used to perform all data analyses, generate tables, figures, and listings. | |
| Reporting Area | |
| HARP Server | : US1SALX00259 |
| HARP Area | : \arprod\gsk2798745\mid201881\final_01 |
| QC Spreadsheet | : \arprod\gsk2798745\mid201881\final_01\documents |
| Analysis Datasets | |
| Analysis datasets will be created according to Integrated Data Standards Library standards. | |

### **Reporting Standards**

### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses :
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
- Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables or figures, unless otherwise stated.
- All unscheduled visits will be listed.

### **Descriptive Summary Statistics**

| • | |
|------------------|--------------------------------------------|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |

| Reporting of Pharmacokinetic Concentration | |
|---|---|
| Descriptive Summary | Refer to IDSL Statistical Principle 6.06.1 |
| Statistics | Assign zero NQ values (Refer to GUI_51487 for further details) |
| Reporting of Pharma | cokinetic Parameters |
| Descriptive Summary<br>Statistics (Log<br>Transformed Data) | N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data and between geometric coefficient of variation (CV <sub>b/w</sub> (%)): $ \text{CV}_{\text{b}} \text{ (\%)} = \sqrt{\left(\text{exp}(\text{SD}^2) - 1\right) * 100} $ |
| | (NOTE: SD is the SD of log transformed data) |
| Parameters Not | tmax, first point, last point and number of points used in the determination |
| Being Log | of Lambda_λz. |
| Transformed | |
| Parameters Not | tmax, first point, last point and number of points used in the determination |
| Being Summarised | of Lambda_λz. |
| Listings | Include the first point, last point and number of points used in the |
| | determination of Lambda_λz. |
| Graphical Displays | |
| Refer to IDSL Statistical Principles 7.01 to 7.13. | |

### 11.5. Appendix 5: Derived and Transformed Data

### 11.5.1. General

### Multiple Measurements at One Time Point

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- For DLco standard practice is to attempt three measures. A pulmonologist will indicate
  which of the three measures are valid, and then a mean will be taken of all valid measures
  to be used as the measurement for that time point. If there is only one valid measure, that
  measure will be used.

### **Study Day**

- Calculated as the number of days from randomisation date:
  - [1] Ref Date = Missing  $\rightarrow$  Study Day = Missing
  - [2] Ref Date < Randomisation Date → Study Day = Ref Date Randomisation Date
  - [3] Ref Data ≥ Randomisation Date → Study Day = Ref Date (Randomisation Date) + 1

### 11.5.2. Study Population

### **Demographics**

### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - [1] Any subject with a missing day will have this imputed as day '15'.
  - [2] Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

### **Body Mass Index (BMI)**

• Calculated as Weight (kg) / [Height (m)]<sup>2</sup>

### **Extent of Exposure**

 Number of days of exposure to study drug will be calculated using dates from the trial medication form. The duration of exposure in days will be based on the formula:

### **Duration of Exposure in Days = Treatment Stop Date – (Start Date + 1)**

 Subjects who were randomized but did not report a treatment start date will be categorized as having zero days of exposure. The cumulative dose will be based on the formula:

### **Cumulative Dose = Sum of (Number of Days x Total Daily Dose)**

 If there are any treatment breaks during the study, then the exposure data will be adjusted accordingly.

### 11.5.3. Safety

### +++ ECG Parameters +++

### **RR Interval**

- IF RR interval (msec) is not provided directly, then RR can be derived as :
  - o If QTcB is machine read & QTcF is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

o If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^3 \right] * 1000$$

 If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value THEN do not derive.

### Corrected QT Intervals

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fredericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTCF will be derived as :

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

### +++ Laboratory Parameters +++

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1.
- If there is more than one value of a particular parameter for a subject for a visit, the scheduled value will be used in summary; all values will be listed.

# 11.6. Appendix 6: Premature Withdrawals & Handling of Missing Data

## 11.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Subject study completion was defined as Safety who either prematurely withdrawn or completed FU visits and assessments. |
| | Withdrawn subjects were not replaced in the study. |
| | <ul> <li>All available data from subjects who were withdrawn from the study will be listed<br/>and all available planned data will be included in summary tables and figures,<br/>unless otherwise specified.</li> </ul> |

## 11.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank<br/>fields on the collection instrument:</li> </ul> |
| | <ul><li>[1] These data will be indicated by the use of a "blank" in subject listing displays.</li><li>[2] Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li></ul> |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

## 11.6.2.1. Handling of Missing Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: |
| | <ul> <li>For a missing start day, the 1st of the month will be used unless this is before the start date of investigational product; in this case the study treatment start date will be used (and hence the event is considered Ontreatment as per Section 11.3 Appendix 1: Treatment States and Phases.</li> <li>For a missing stop day, the last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> |
| | Start or end dates which are completely missing (i.e. no year specified) will |

| Element | Reporting Detail |
|---------|---------------------------------------------|
| | remain missing, with no imputation applied. |

## 11.6.2.2. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant Medications | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be<br/>imputed using the following convention:</li> </ul> |
| | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> <li>The recorded partial date will be displayed in listings.</li> </ul> |
| Adverse<br>Events | <ul> <li>Any partial dates for adverse events will be raised to data management. If the<br/>full date cannot be ascertained, the following assumptions will be made:</li> </ul> |
| | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month.</li> <li>However, if these results in a date prior to Week 1 Day 1 and the event could possibly have occurred during treatment from the partial information, then the Week 1 Day 1 date will be assumed to be the start date.</li> <li>The AE will then be considered to start on-treatment (worst case).</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 11.7. Appendix 7: Values of Potential Clinical Importance

## 11.7.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | | Male | | 0.54 |
| Hematocrit | Ratio of 1 | Female | | 0.54 |
| | | $\Delta$ from BL | ↓0.075 | |
| | | Male | | 180 |
| Hemoglobin | g/L | Female | | 180 |
| | | $\Delta$ from BL | ↓25 | |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.8 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | mmol/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | mmol/L | $\Delta$ from BL | | ↑ 44.2 |
| Glucose | mmol/L | | 3 | 9 |
| Magnesium | mmol/L | | 0.5 | 1.23 |
| Phosphorus | mmol/L | | 0.8 | 1.6 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| Total CO2 | mmol/L | | 18 | 32 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5xULN |
| | µmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |

## 11.7.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|----------------------------|-------|------------------------|-------|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | msec | > 450 | |
| Absolute PR Interval | msec | < 110 | > 220 |
| Absolute QRS Interval | msec | < 75 | > 110 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | > 60 | |

# 11.7.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

## 11.8. Appendix 8: Laboratory A&R Dataset Details

| | Norm. | | al Range | Anticipated Direction of | |
|---|---|---|---|---|---|
| Panel [1] | Parameter | Unit | Low High | | Change with Treatment |
| | Serum Albumin | G/L | 32 | 50 | |
| | Alkaline Phosphatase | IU/L | 20 | 125 | |
| | ALT | IU/L | 0 | 48 | 1 |
| | AST | IU/L | 0 | 42 | 1 |
| | BUN (UREA) | MMOL/L | 2.5 | 10.5 | |
| | Calcium | MMOL/L | 2.12 | 2.56 | |
| | Chloride | MMOL/L | 95 | 108 | |
| | Creatinine | UMOL/L | 67.2 | 129.1 | Safety laboratory |
| Fasted Chemistry | Creatinine Clearance | N/A | N/A | N/A | parameters not expected |
| | Direct Bilirubin | UMOL/L | 0 | 6 | to change |
| | GGT | IU/L | 0 | 75 | |
| | Glucose, fasting | MMOL/L | 3.9 | 5.5 | |
| | Potassium | MMOL/L | 3.5 | 5.3 | |
| | Sodium | MMOL/L | 135 | 146 | |
| | Total Bilirubin | UMOL/L | 0 | 22 | |
| | Total Protein | G/L | 60 | 85 | |
| | Uric Acid | UMOL/L | 240 | 510 | |
| | HDL | MMOL/L | 0.9 | 99.99 | Safety laboratory |
| 1 | LDL (Calculated) | MMOL/L | 0 | 3.35 | parameters not expected |
| Lipid | Total Cholesterol | MMOL/L | 0 | 5.15 | to change |
| | Triglycerides | MMOL/L | 0 | 2.24 | |
| | Blood | Dipstick | N/AP | N/AP | |
| | Bacteria | Microy | N/AP | N/AP | |
| | Hyaline Casts (N/A) | N/A | N/AP | N/AP | Not able to specify |
| Urinalysis | Nitrite | Dipstick | N/AP | N/AP | specifically. |
| | Protein | Dipstick | N/AP | N/AP | |
| | RBC | Microscopy | N/AP | N/AP | |
| | Specific Gravity | N/A | N/AP | N/AP | |
| | WBC | GI/L | 3.8 | 10.8 | |
| | Basophils | GI/L | 0 | 0.2 | |
| | Eosinophils | GI/L | 0.05 | 0.55 | |
| | Hemoglobin | G/L | 118 | 168 | |
| Haematology | Hematocrit | 1 | 0.41 | 0.5 | |
| | Lymphocytes | GI/L | 0.85 | 4.1 | Safety laboratory |
| | MCV | FL | 82 | 103 | parameters not expected |
| | MCH | PG | 27 | 33 | to change |
| | MCHC | G/L | 320 | 360 | |
| | Monocytes | GI/L | 0.2 | 1.1 | |
| | Neutrophils | GI/L | 130 | 400 | |
| | Platelet Count | GI/L | 130 | 400 | |
| | RBC Count | TI/L | 3.7 | 5.5 | |
| | WBC Count (Absolute) | GI/L | 3.8 | 10.8 | |

## NOTE:

- N/A = Not available on DM dataset during RAP completion.
- N/AP = No ranges are normally provided for parameters.

## 11.9. Appendix 9: Biomarker A&R Dataset Details

| Parameters (BICATCD Code) | Sample | Unit | LLQ | ULQ |
|---|---|---|---|---|
| Dataset : Biomark (QUEST) | | | | |
| Adiponectin (ADPN) | Serum | MG/L | 2 | 61 |
| Albumin (ALB) | Urine | MG/L | 3 | 9999 |
| Creatinine (CREAT) | Urine | MMOL/L | 0.2 | 999999.9 |
| C-peptide (MMT) (CPEP) | Serum | NMOL/L | 0.1 | 9999.99 |
| C-Reactive Protein, Highly Sensitive (CRPHS) | Serum | MG/L | 0.3. | 800 |
| CXCL10 / IP-10 (IP10) | Serum | NG/L | 54.5 | 56000 |
| Fructosamine (FRUC) | Serum | UMOL/L | 20 | 1000 |
| Glucose (MMT) (GLUC) | Plasma | MMOL/L | 1.1 | 277.5 |
| Glucagon (MMT) (No data for IA) | Plasma | N/A | N/A | N/A |
| Glycohemoglobin A1c (HbA1c) | Whole<br>Blood | MMOL/L | 3 | 18.9 |
| Highly Sensitive Interleukin-6 (IL-6) | Serum | NG/L | 0.156 | 640 |
| Insulin (MMT) (INS) | Serum | PMOL/L | 12 | 99999 |
| Intercellular Adhesion Molecule, Soluble (sICAM) | Serum | NG/L | 312 | 3200000 |
| Matrix Metalloproteinase-9 (MMP-9) | Serum | NG/L | 975 | 40000000 |
| Non-Esterified Fatty Acids (NEFA) | Serum | MMOL/L | 0.03 | 9 |
| Monocyte Chemotactic protein-1 (MCP1) | Urine | NG/L | 3.12 | 800 |
| Plasminogen Activator Inhibitor-1 (PAI-1) | Plasma | NG/L | 153 | 20000000 |
| Resistin (RESIST) | Serum | MCG/L | 0.8 | 800 |
| Dataset : IMGEN (GSK Clinical Immunology) | | | | |
| Interleukin 18 – Complex (IL18C) | Serum | pg/mL | 19.5 | N/AP |
| Interleukin 18 – Free (IL8F) | Serum | pg/mL | 4 | N/AP |

### NOTE:

- Urine biomarkers will be reported as ratios to creatinine i.e. Albumin/creatinine (ACR) and MCP-1/creatinine.
- N/A Not available on DM dataset during RAP completion.
- N/AP = No ranges are normally provided for parameters.
# 11.10. Appendix 10 – Abbreviations & Trade Marks

#### 11.10.1. Abbreviations

| Abbreviation | Description |
|---|---|
| AE | Adverse Event |
| GSK | GlaxoSmithKline |
| AE | Adverse Event |
| ALT | Alanine aminotransferase (SGPT) |
| AST | Aspartate aminotransferase (SGOT) |
| AUC | Area under concentration-time curve |
| AUC(0-∞) | Area under the concentration-time curve from time zero (pre-dose) |
| | extrapolated to infinite time |
| BMI | Body mass index |
| BPM | Beat Per Minute |
| BQL | Below the quantification limit |
| CL | Systemic clearance of parent drug |
| Cmax | Maximum observed concentration |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CPSR | Clinical Pharmacology Study Report |
| CS | Clinical Statistics |
| CPSSO | Clinical Pharmacology Science and Study Operations |
| CV | Coefficient of variance |
| DM | Data Management |
| FPG | Fasting Plasma Glucose |
| GSK | GlaxoSmithKline |
| HOMA-%B | Homeostasis Model Assessment (β-cell function) |
| HOMA-%S | Homeostasis Model Assessment (Insulin sensitivity) |
| HR | Heart rate |
| ICH | International Conference on Harmonization of Technical Requirements |
| | for Registration of Pharmaceuticals for Human Use |
| IDSL | Integrated Data Standards Library |
| IL | Interleukin |
| Kg | Kilogram |
| $\lambda z$ | Terminal phase rate constant |
| LLQ | Lower limit of quantification |
| MMRM | Mixed models repeated measures |
| MMT | Mixed Meal Test |
| msec | Milliseconds |
| NQ | Non-quantifiable concentration measured as below LLQ |
| OB | Obese |
| PK | Pharmacokinetic |
| QC | Quality control |
| QTc | QT duration corrected |

| Abbreviation | Description |
|---|---|
| QTcB | QT duration corrected for heart rate by Bazett's formula |
| QTcF | QT duration corrected for heart rate by Fridericia's formula |
| RAP | Reporting and Analysis Plan |
| RNA | Ribonucleic acid |
| SAS | Statistical Analysis Software |
| SI | System Independent |
| STAT | Signal tranducer and activator of transcription |
| SD | Standard deviation |
| SOP | Standard Operating Procedure |
| T | Infusion duration |
| t OR tlast | Time of last observed quantifiable concentration |
| t½ | Terminal phase half-life |
| τ | Dosing interval |
| tlag | Lag time before observation of drug concentrations in sampled matrix |
| tmax | Time of occurrence of Cmax |
| TNF-α | Tumour necrosis factor – alpha |
| ULQ | Upper limit of quantification |
| ULN | Upper limit of normal |
| UK | United Kingdom |
| VAS | Visual analogue score |
| Vss | Volume of distribution at steady state |
| WBA | Whole blood assay |
| WBC | White blood cells |

#### 11.10.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies | |
|---------------------------------------------------------|---|
| NONE | 1 |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| NONMEM |
| SAS |
| WinNonlin |

#### 11.13. Appendix 11: List of Data Displays

#### 11.13.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|---------------|--------------|
| Study Population | 1.01 to 1.11 | N/A |
| Efficacy | 2.01 to 2.32 | 2.01 to 2.72 |
| Safety | 3.01 to 3.21 | N/A |
| Pharmacokinetic | 4.01 to 4.05 | 4.01 to 4.02 |
| Section | Listings | |
| ICH Listings | tings 1 to 23 | |
| Other Listings | 24 t | o 41 |

The numbering of the TLF's below is a suggestion and can be altered by the programmers if needed. If the programmers need to change the numbering, please add new numbers to the end of the sequence.

#### 11.13.2. Deliverable [Priority]

| Delivery Priority <sup>1</sup> | Description |
|---|---|
| IA | "Interim" Analysis Part A (after completion of approximately 6 patients) |
| SAC 2 | Part A Final Statistical Analysis Complete |

#### 11.13.3. Mock Example Numbering

Non IDSL specifications will be referred as detailed below and where appropriate an example mock-up table is provided in Appendix 12:

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |

#### NOTE:

 Non-Standard displays are indicated in the IDSL / TST ID / Example Shell' or Programming Notes' column as '[Non-Standard] + Reference.'

# 11.13.4. Study Population Tables

| Study I | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.01 | All Subjects | ES1 | Summary of Subject Disposition | | SAC [2] |
| 1.02 | Screening<br>Population | ES6 | Summary of Reasons for Screening Failure | | SAC [2] |
| 1.03 | All Subjects | ES5 | Summary of Reasons for Withdrawals | | SAC [2] |
| 1.04 | All Subjects | DV1a | Summary of Important Protocol Deviations | | SAC [2] |
| 1.05 | All Subjects | SA2 | Summary of Deviations Leading to Exclusion from Per Protocol Population | | SAC [2] |
| Demog | raphics | | | | |
| 1.06 | All Subjects | DM1 | Summary of Demographic Characteristics | Make twice, pooled and by site | IA, SAC [2] |
| 1.07 | All Subjects | DM5 | Summary of Race and Racial Combinations | Make twice, pooled and by site | SAC [2] |
| 1.08 | Enrolled | DM11 | Summary of Age Ranges | | SAC [2] |
| 1.12 | Enrolled | NS1 | Summary of Number of Subjected by Country and Site ID | | SAC[2] |
| 1.09 | All Subjects | SA1 | Summary of Study Populations | | SAC [2] |
| Medica | Medical Condition & Con Meds | | | | |
| 1.10 | All Subjects | MH1 | Summary of [Current/Past] Medical Conditions | Make twice, pooled and by site | SAC [2] |

#### CONFIDENTIAL

| Study Population Tables | | | | | |
|---|---|---|---|---|---|
| No. Population IDSL / TST ID / Example Shell Title Programming Notes | | | | | Deliverable<br>[Priority] |
| 1.11 | All Subjects | CM1 | Summary of Most Frequently used Concomitant Medications by Generic Term | Footnote: Most Frequently means the overall concomitant medication used is >= 10% | SAC [2] |

# 11.13.5. Efficacy Tables

| Efficac | y Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| DLco | | | | | |
| 2.01 | Analysis | Non-Standard<br>EFF_T1 | Summary Statistics of DLco | DLco has measures on Baseline, Day 4, 5, and 7 for each treatment period and follow-up. Create this table twice, one table with only Mayo patients and another table with only Hennepin patients | IA, SAC [2] |
| 2.02 | Analysis | Non-Standard<br>EFF_T2 | Summary Statistics of DLco Change from Baseline | Create this table twice, one table with only Mayo patients and another table with only Hennepin patients | IA, SAC [2] |
| 2.03 | Analysis | Non-Standard<br>EFF_T12 | Summary Statistics of DLco Change from Intervention | Create this table twice, one table with only Mayo patients and another table with only Hennepin patients. This should be the Mean and SD of the Post-Pre difference. | IA, SAC [2] |
| 2.04 | Analysis | Non-Standard<br>EFF_T6 | Summary of Statistical Analysis Results of DLco | Models should be run with only Mayo patients. Hennepin patients are excluded because of methodological differences. | IA, SAC [2] |
| Alveola | ar-capillary Co | nductance (D <sub>M</sub> ) | | | |
| 2.05 | Analysis | Non-Standard<br>EFF_T3 | Summary Statistics of Gas Transfer Tests | DLno, Dm, Vc, and Dm/Vc have measures on<br>Baseline, Day 4, 5, and 7 for each treatment period<br>and follow-up | SAC [2] |
| 2.06 | Analysis | Non-Standard<br>EFF_T2 | Summary Statistics of Gas Transfer Tests Change from Baseline | DLno, Dm, Vc, and Dm/Vc have measures on Baseline, Day 4, 5, and 7 for each treatment period and follow-up. Baseline is day -1 for exercise and chronic values, but should be calculated as post minus pre for Saline. | SAC [2] |

| Efficac | y Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.07 | Analysis | Non-Standard<br>EFF_T12 | Summary Statistics of Gas Transfer Tests Change from Intervention | DLno, Dm, Vc, and Dm/Vc have measures on Baseline and Day 5 and 7 for each treatment period. This should be the Mean and SD of the Post-Pre difference. | IA, SAC [2] |
| Ventila | tory Efficiency | / | | | |
| 2.08 | Analysis | Non-Standard<br>EFF_T7 | Summary Statistics of VE/VCO <sub>2</sub> Ratio | VE/VCO <sub>2</sub> ratio has measures on Baseline and Day 7 before and after 3-minutes step test. Create this table twice, one table with all patients and another table with Hennepin patients excluded from the statistics. | SAC [2] |
| 2.09 | Analysis | Non-Standard<br>EFF_T8 | Summary Statistics of VE/VCO <sub>2</sub> Ratio Change from Baseline | VE/VCO <sub>2</sub> ratio has measures on Baseline and Day 7 before and after 3-minutes step test. Create this table twice, one table with all patients and another table with Hennepin patients excluded from the statistics. | SAC [2] |
| Pulmor | nary Function | | | | |
| 2.10 | Analysis | Non-Standard<br>EFF_T4 | Summary Statistics of Pulmonary Function Tests | Pulmonary function (FVC, FEV <sub>1</sub> , FEF <sub>25-75</sub> , FEF <sub>50</sub> , FEF <sub>75</sub> ) has measures on Baseline, Day 4 and Day 7 for each treatment period. Pool all patients. | SAC [2] |
| 2.11 | Analysis | Non-Standard<br>EFF_T5 | Summary Statistics of Pulmonary Function Tests<br>Change from Baseline | Pulmonary function (FVC, FEV <sub>1</sub> , FEF <sub>25-75</sub> , FEF <sub>50</sub> , FEF <sub>75</sub> ) has measures on Baseline, Day 4, and Day 7 for each treatment period. Pool all patients. | SAC [2] |
| 2.12 | Analysis | Non-Standard<br>EFF_T4 | Summary Statistics of Pulmonary Function Tests by Site | Pulmonary function (FVC, FEV <sub>1</sub> , FEF <sub>25-75</sub> , FEF <sub>50</sub> , FEF <sub>75</sub> ) has measures on Baseline, Day 4 and Day 7 for each treatment period. Create this table twice, one table with Mayo patients and another table with Hennepin patients. | SAC [2] |

| Efficac | y Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.13 | Analysis | Non-Standard<br>EFF_T5 | Summary Statistics of Pulmonary Function Tests<br>Change from Baseline by Site | Pulmonary function (FVC, FEV <sub>1</sub> , FEF <sub>25-75</sub> , FEF <sub>50</sub> , FEF <sub>75</sub> ) has measures on Baseline, Day 4, and Day 7 for each treatment period. Create this table twice, one table with Mayo patients and another table with Hennepin patients. | SAC [2] |
| Dyspne | ea | | | | |
| 2.14 | Analysis | Non-Standard<br>EFF_T9 | Summary Statistics Dyspnea Score | Dyspnea Score has measures at Baseline pre and post exercise, Day 5 pre-saline sitting and supine, Day 7 pre and post exercise for each treatment period and at follow-up pre and post exercise | SAC [2] |
| 2.15 | Analysis | Non-Standard<br>EFF_T5 | Summary Statistics Change from Baseline Dyspnea<br>Score | Dyspnea Score change from baseline has measures at Baseline post exercise, Day 5 pre-saline sitting and supine, Day 7 pre and post exercise for each treatment period and at follow-up pre and post exercise | SAC [2] |
| SF-36 s | score | l | | | |
| 2.16 | Analysis | SF2 | Summary Statistics SF-36 Score | SF-36 Score has measures at Baseline and Day 7 for each treatment period and follow-up. Add additional rows for questions 3a to 3j to be looked at along with the domain scores | SAC [2] |
| 2.17 | Analysis | SF4 | Summary Statistics of Change from Baseline SF-36<br>Score | SF-36 Score change from Baseline has a measure at Day 7 for each treatment period and follow-up. Add additional rows for questions 3a to 3j to be looked at along with the domain scores | SAC [2] |

| Efficac | Efficacy Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Tropon | in | | | | |
| 2.18 | All Subject | LB1 | Summary Statistics of Troponin | | SAC [2] |
| 2.19 | All Subject | LB3 | Summary Statistics of Troponin Change from Baseline | | SAC [2] |
| Respira | Respiratory Rate | | | | |
| 2.20 | All Subject | EFF_T11 | Summary Statistics of Respiratory Rate | | SAC [2] |

# 11.13.6. Efficacy Figures

| Efficac | Efficacy Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Gas tra | ansfer measure | e | | • | |
| 2.01 | Analysis | Non-Standard<br>EFF_F1 | Spaghetti Plot of DLco | DLco has measures at Baseline, Day 4, Day 5, and Day 7 for each period as well as screening and follow-up. Includes pre/post exercise and saline challenge. | SAC [2] |
| 2.02 | Analysis | Non-Standard<br>EFF_F22 | Spaghetti Plot of DLco by Site | DLco has measures at Baseline, Day 4, Day 5, and Day 7 for each period. Excludes post exercise and post saline challenge. | SAC [2] |
| 2.03 | Analysis | Non-Standard<br>EFF_F2 | Mean (95% CI) Plot of DLco | Create this graph twice, one graph with Mayo patients and another graph with Hennepin patients | SAC [2] |
| 2.04 | Analysis | Non-Standard<br>EFF_F3 | Mean (95% CI) Plot of Chronic DLco | Create this graph twice, one graph with Mayo patients and another graph with Hennepin patients | SAC [2] |
| 2.05 | Analysis | Non-Standard<br>EFF_F4 | Plot of DLco by Individual and Treatment | DLco has measures at Baseline, Day 4, Day 5, and Day 7 for each treatment as well as screening and follow-up. Includes pre/post exercise and saline challenge. Horizontal line represents baseline values | SAC [2] |
| 2.06 | Analysis | Non-Standard<br>EFF_F5 | Plot of Change from Baseline for Chronic DLco by Individual and Treatment | Only pre-challenge DLco values | SAC [2] |

| Efficac | Efficacy Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.07 | Analysis | Non-Standard<br>EFF_F6 | Mean (95% CI) Plot of DLco Change from Baseline | DLco has means at Baseline, Day 4, Day 5, and Day 7 for each treatment and includes pre/post exercise and saline challenge. Baseline is minus day -1 for exercise and no challenge, but should be calculated as post minus pre for Saline. Create this graph twice, one graph with Mayo patients and another graph with Hennepin patients | SAC [2] |
| 2.08 | Analysis | Non-Standard<br>EFF_F7 | Mean (95% CI) Plot of Exercise DLco | DLco has measures at Baseline and Day 7 for each treatment and a follow-up. Graph should include pre/post exercise values. Create this graph twice, one graph with Mayo patients and another graph with Hennepin patients | SAC [2] |
| 2.09 | Analysis | Non-Standard<br>EFF_F8 | Mean (95% CI) Plot of Change from Exercise for DLco | DLco has means at Baseline and Day 7 for each treatment and a follow-up. The bars represent the mean change from just prior to exercise to post exercise. mean(Post-Pre) Create this graph twice, one graph with Mayo patients and another graph with Hennepin patients | SAC [2] |
| 2.10 | Analysis | Non-Standard<br>EFF_F9 | Mean (95% CI) Plot of Percent Change from Exercise for DLco | DLco has means at Baseline and Day 7 for each treatment and a follow-up. The bars represent the mean percent change from just prior to exercise to post exercise. Create this graph twice, one graph with Mayo patients and another graph with Hennepin patients | SAC [2] |

| Efficac | Efficacy Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.11 | Analysis | Non-Standard<br>EFF_F10 | Mean (95% CI) Plot of Percent Change from Saline for DLco | DLco has means at Day 5 for each treatment and a follow-up. The bars represent the mean percent change from just prior to exercise to post saline infusion. Create this graph twice, one graph with Mayo patients and another graph with Hennepin patients | SAC [2] |
| 2.12 | Analysis | Non-Standard<br>EFF_F24 | Bar Plot of Saline Challenge for DLco by Subject | Bars should be able to distinguish pre- and post-<br>saline values. On the bars for each patient should be<br>text. The text is the difference between before and<br>after and the percent change, as seen in the mock up<br>Create this graph twice, one graph with Mayo<br>patients and another graph with Hennepin patients | SAC [2] |
| 2.13 | Analysis | Non-Standard<br>EFF_F1 | Spaghetti Plot of DLno | DLno has measures at Baseline, Day 4, Day 5, and Day 7 for each period as well as screening and follow-up. Includes pre/post exercise and saline challenge. | SAC [2] |
| 2.14 | Analysis | Non-Standard<br>EFF_F2 | Mean (95% CI) Plot of DLno | | SAC [2] |
| 2.15 | Analysis | Non-Standard<br>EFF_F3 | Mean (95% CI) Plot of Chronic DLno | | SAC [2] |
| 2.16 | Analysis | Non-Standard<br>EFF_F4 | Plot of DLno by Individual and Treatment | DLno has measures at Baseline, Day 4, Day 5, and Day 7 for each treatment as well as screening and follow-up. Includes pre/post exercise and saline challenge. Horizontal line represents baseline values | SAC [2] |
| 2.17 | Analysis | Non-Standard<br>EFF_F5 | Plot of Change from Baseline for Chronic DLno by Individual and Treatment | Only pre-challenge DLno values | SAC [2] |

| Efficac | Efficacy Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.18 | Analysis | Non-Standard<br>EFF_F6 | Mean (95% CI) Plot of DLno Change from Baseline | DLno has means at Baseline, Day 4, Day 5, and Day 7 for each treatment and includes pre/post exercise and saline challenge. Baseline is minus day -1 for exercise and no challenge, but should be calculated as post minus pre for Saline. | SAC [2] |
| 2.19 | Analysis | Non-Standard<br>EFF_F7 | Mean (95% CI) Plot of Exercise DLno | DLno has measures at Baseline and Day 7 for each treatment and a follow-up. Graph should include pre/post exercise values. | SAC [2] |
| 2.20 | Analysis | Non-Standard<br>EFF_F8 | Mean (95% CI) Plot of Change from Exercise for DLno | DLno has means at Baseline and Day 7 for each treatment and a follow-up. The bars represent the mean change from just prior to exercise to post exercise. mean(Post-Pre) | SAC [2] |
| 2.21 | Analysis | Non-Standard<br>EFF_F9 | Mean (95% CI) Plot of Percent Change from Exercise for DLno | DLno has means at Baseline and Day 7 for each treatment and a follow-up. The bars represent the mean percent change from just prior to exercise to post exercise. | SAC [2] |
| 2.22 | Analysis | Non-Standard<br>EFF_F10 | Mean (95% CI) Plot of Percent Change from Saline for DLno | DLno has means at Day 5 for each treatment and a follow-up. The bars represent the mean percent change from just prior to exercise to post saline infusion. | SAC [2] |
| 2.23 | Analysis | Non-Standard<br>EFF_F24 | Bar Plot of Saline Challenge for DLno by Subject | Bars should be able to distinguish pre- and post-<br>saline values. On the bars for each patient should be<br>text. The text is the difference between before and<br>after and the percent change, as seen in the mock up<br>Create this graph twice, one graph with Mayo<br>patients and another graph with Hennepin patients | SAC [2] |
| 2.24 | Analysis | Non-Standard<br>EFF_F1 | Spaghetti Plot of D <sub>M</sub> | D <sub>M</sub> has measures at Baseline, Day 4, Day 5, and Day 7 for each period as well as screening and follow-up. Includes pre/post exercise and saline challenge. | SAC [2] |

| Efficac | Efficacy Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.25 | Analysis | Non-Standard<br>EFF_F2 | Mean (95% CI) Plot of D <sub>M</sub> | | SAC [2] |
| 2.26 | Analysis | Non-Standard<br>EFF_F3 | Mean (95% CI) Plot of Chronic D <sub>M</sub> | | SAC [2] |
| 2.27 | Analysis | Non-Standard<br>EFF_F4 | Plot of D <sub>M</sub> by Individual and Treatment | D <sub>M</sub> has measures at Baseline, Day 4, Day 5, and Day 7 for each treatment as well as screening and follow-up. Includes pre/post exercise and saline challenge. Horizontal line represents baseline values | SAC [2] |
| 2.28 | Analysis | Non-Standard<br>EFF_F5 | Plot of Change from Baseline for Chronic D <sub>M</sub> by Individual and Treatment | Only pre-challenge D <sub>M</sub> values | SAC [2] |
| 2.29 | Analysis | Non-Standard<br>EFF_F6 | Mean (95% CI) Plot of D <sub>M</sub> Change from Baseline | D <sub>M</sub> has means at Baseline, Day 4, Day 5, and Day 7 for each treatment and includes pre/post exercise and saline challenge. Baseline is minus day -1 for exercise and no challenge, but should be calculated as post minus pre for Saline. | SAC [2] |
| 2.30 | Analysis | Non-Standard<br>EFF_F7 | Mean (95% CI) Plot of Exercise D <sub>M</sub> | D <sub>M</sub> has measures at Baseline and Day 7 for each treatment and a follow-up. Graph should include pre/post exercise values. | SAC [2] |
| 2.31 | Analysis | Non-Standard<br>EFF_F8 | Mean (95% CI) Plot of Change from Exercise for D <sub>M</sub> | D <sub>M</sub> has means at Baseline and Day 7 for each treatment and a follow-up. The bars represent the mean change from just prior to exercise to post exercise. mean(Post-Pre) | SAC [2] |
| 2.32 | Analysis | Non-Standard<br>EFF_F9 | Mean (95% CI) Plot of Percent Change from Exercise for $D_M$ | D <sub>M</sub> has means at Baseline and Day 7 for each treatment and a follow-up. The bars represent the mean percent change from just prior to exercise to post exercise. | SAC [2] |

| Efficac | Efficacy Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.33 | Analysis | Non-Standard<br>EFF_F10 | Mean (95% CI) Plot of Percent Change from Saline for $D_M$ | D <sub>M</sub> has means at Day 5 for each treatment and a follow-up. The bars represent the mean percent change from just prior to exercise to post saline infusion. | SAC [2] |
| 2.34 | Analysis | Non-Standard<br>EFF_F1 | Spaghetti Plot of Vc | Vc has measures at Baseline, Day 4, Day 5, and Day 7 for each period as well as screening and follow-up. Includes pre/post exercise and saline challenge. | SAC [2] |
| 2.35 | Analysis | Non-Standard<br>EFF_F2 | Mean (95% CI) Plot of Vc | | SAC [2] |
| 2.36 | Analysis | Non-Standard<br>EFF_F3 | Mean (95% CI) Plot of Chronic Vc | | SAC [2] |
| 2.37 | Analysis | Non-Standard<br>EFF_F4 | Plot of Vc by Individual and Treatment | Vc has measures at Baseline, Day 4, Day 5, and Day 7 for each treatment as well as screening and follow-up. Includes pre/post exercise and saline challenge. Horizontal line represents baseline values | SAC [2] |
| 2.38 | Analysis | Non-Standard<br>EFF_F5 | Plot of Change from Baseline for Chronic Vc by Individual and Treatment | Only pre-challenge Vc values | SAC [2] |
| 2.39 | Analysis | Non-Standard<br>EFF_F6 | Mean (95% CI) Plot of Vc Change from Baseline | Vc has means at Baseline, Day 4, Day 5, and Day 7 for each treatment and includes pre/post exercise and saline challenge. Baseline is minus day -1 for exercise and no challenge, but should be calculated as post minus pre for Saline. | SAC [2] |
| 2.40 | Analysis | Non-Standard<br>EFF_F7 | Mean (95% CI) Plot of Exercise Vc | Vc has measures at Baseline and Day 7 for each treatment and a follow-up. Graph should include pre/post exercise values. | SAC [2] |

| Efficac | y Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.41 | Analysis | Non-Standard<br>EFF_F8 | Mean (95% CI) Plot of Change from Exercise for Vc | Vc has means at Baseline and Day 7 for each treatment and a follow-up. The bars represent the mean change from just prior to exercise to post exercise. mean(Post-Pre) | SAC [2] |
| 2.42 | Analysis | Non-Standard<br>EFF_F23 | Forest Plot of DL End Points Change | Forest plot of Dlco, Dlno, Vc, and Dm change from baseline to day 7, change from pre and post saline for Dlco and change from pre/post exercise on day 7 for Dlco. Include the mean absolute change next to the box plot as seen in the mock-up | SAC[2] |
| 2.43 | Analysis | Non-Standard<br>EFF_F9 | Mean (95% CI) Plot of Percent Change from Exercise for Vc | Vc has means at Baseline and Day 7 for each treatment and a follow-up. The bars represent the mean percent change from just prior to exercise to post exercise. | SAC [2] |
| 2.44 | Analysis | Non-Standard<br>EFF_F10 | Mean (95% CI) Plot of Percent Change from Saline for Vc | Vc has means at Day 5 for each treatment and a follow-up. The bars represent the mean percent change from just prior to exercise to post saline infusion. | SAC [2] |
| Ventila | atory Efficienc | у | | | |
| 2.45- | Analysis | Non-Standard<br>EFF_F11 | Plot of VE/VCO <sub>2</sub> | Has 5 measures at Baseline, Day 7, and Follow-Up | SAC[2] |
| 2.46 | Analysis | Non-Standard<br>EFF_F12 | Mean (95% CI) Plot of VE/VCO <sub>2</sub> | Has means for each of the 5 measures at baseline,<br>Day 7 and Follow-Up | SAC[2] |
| 2.47 | Analysis | Non-Standard<br>EFF_F13 | Plot of VE/VCO₂ Change from Day -1 | Is the difference between day -1 and day 7 for each time point in the exercise test (e.g. at rest day 7 – at rest day -1, post 1 min day 7 - post 1 min day -1) | SAC[2] |

| Efficac | Efficacy Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.48 | Analysis | Non-Standard<br>EFF_F14 | Mean (95% CI) Change from Baseline Plot of VE/VCO <sub>2</sub> | Mean values of the points calculated for previous plot | SAC[2] |
| 2.49 | Analysis | Non-Standard<br>EFF_F15 | Plot of VE/VCO <sub>2</sub> Change from Rest | Has 5 measures at baseline and Day 7 for each treatment along a with follow-up. Bars represent the difference the time measure and rest within a day and treatment. The number is the difference between the active and placebo bars. | SAC[2] |
| 2.50 | Analysis | Non-Standard<br>EFF_F16 | Mean (95% CI) Plot of VE/VCO₂ Change from Rest | Has means at Day 7 | SAC[2] |
| Pulmo | nary Function | | | | |
| 2.51 | Analysis | Non-Standard<br>EFF_F17 | Spaghetti Plot of FVC | FVC has means at Baseline, Day 4 and Day 7 for each treatment and a follow-up measure | SAC[2] |
| 2.52 | Analysis | Non-Standard<br>EFF_F18 | Mean (95% CI) Plot of FVC | FVC has means at Baseline, Day 4 and Day 7 for each treatment and a follow-up measure | SAC[2] |
| 2.53 | Analysis | Non-Standard<br>EFF_F19 | Mean (95% CI) Plot of FVC Change from Baseline | FVC has means at Day 4 and Day 7 | SAC[2] |
| 2.54 | Analysis | Non-Standard<br>EFF_F17 | Spaghetti Plot of FEV <sub>1</sub> | FEV <sub>1</sub> has means at Baseline, Day 4 and Day 7 for each treatment and a follow-up measure | SAC[2] |
| 2.55 | Analysis | Non-Standard<br>EFF_F18 | Mean (95% CI) Plot of FEV <sub>1</sub> | FEV <sub>1</sub> has means at Baseline, Day 4 and Day 7 for each treatment and a follow-up measure | SAC[2] |

| Efficac | Efficacy Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.56 | Analysis | Non-Standard<br>EFF_F19 | Mean (95% CI) Plot of FEV₁ Change from Baseline | FEV₁ has means at Day 4 and Day 7. | SAC[2] |
| 2.57 | Analysis | Non-Standard<br>EFF_F17 | Spaghetti Plot of FEF <sub>25-75</sub> | FEF <sub>25-75</sub> has means at Baseline, Day 4 and Day 7 for each treatment and a follow-up measure | SAC[2] |
| 2.58 | Analysis | Non-Standard<br>EFF_F18 | Mean (95% CI) Plot of FEF <sub>25-75</sub> | FEV <sub>25-75</sub> has means at Baseline, Day 4 and Day 7 for each treatment and a follow-up measure | SAC[2] |
| 2.59 | Analysis | Non-Standard<br>EFF_F19 | Mean (95% CI) Plot of FEF <sub>25-75</sub> Change from Baseline | FEF <sub>25-75</sub> has means at Day 4 and Day 7 | SAC[2] |
| 2.60 | Analysis | Non-Standard<br>EFF_F17 | Spaghetti Plot of FEF <sub>50</sub> | FEF <sub>25-75</sub> has means at Baseline, Day 4 and Day 7 for each treatment and a follow-up measure | SAC[2] |
| 2.61 | Analysis | Non-Standard<br>EFF_F18 | Mean (95% CI) Plot of FEF <sub>50</sub> | FEF <sub>50</sub> has means at Baseline, Day 4 and Day 7 for each treatment and a follow-up measure | SAC[2] |
| 2.62 | Analysis | Non-Standard<br>EFF_F19 | Mean (95% CI) Plot of FEF <sub>50</sub> Change from Baseline | FEF <sub>50</sub> has means at Day 4 and Day 7. | SAC[2] |
| 2.63 | Analysis | Non-Standard<br>EFF_F17 | Spaghetti Plot of FEF <sub>75</sub> | FEF <sub>75</sub> has means at Baseline, Day 4 and Day 7 for each treatment and a follow-up measure | SAC[2] |
| 2.64 | Analysis | Non-Standard<br>EFF_F18 | Mean (95% CI) Plot of FEF <sub>75</sub> | FEF <sub>75</sub> has means at Baseline, Day 4 and Day 7 for each treatment and a follow-up measure | SAC[2] |

| Efficac | y Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.65 | Analysis | Non-Standard<br>EFF_F19 | Mean (95% CI) Plot of FEF <sub>75</sub> Change from Baseline | FEF <sub>75</sub> has means at Day 4 and Day 7. | SAC[2] |
| 2.66 | Analysis | Non-Standard<br>EFF_F23 | Forest Plot of Pulmonary Function Test | Forest plot of FVC, FEV <sub>1</sub> , FEF <sub>25-75</sub> , FEF <sub>50</sub> , FEF <sub>75</sub> . Include the mean absolute change next to the box plot as seen in the mock-up | SAC[2] |
| Dyspn | ea | | | | |
| 2.67 | Analysis | Non-Standard<br>EFF_F17 | Spaghetti Plot of Dyspnea | Dyspnea has measures at Baseline pre and post exercise, Day 5 pre-saline sitting and supine, and Day 7 pre and post exercise | SAC[2] |
| 2.68 | Analysis | Non-Standard<br>EFF_F18 | Mean (95% CI) Plot of Dyspnea | Dyspnea has means at Baseline pre and post exercise, Day 5 pre-saline sitting and supine, and Day 7 pre and post exercise. | SAC[2] |
| 2.69 | Analysis | Non-Standard<br>EFF_F19 | Mean (95% CI) Plot of Dyspnea Change from Baseline | Dyspnea has means at Baseline post exercise, Day 5 pre-saline sitting and supine, and Day 7 pre and post exercise | SAC[2] |
| SF-36 | Score | | | | |
| 2.70 | Analysis | Non-Standard<br>EFF_F19 | Mean (95% CI) Plot of SF-36 Acute Score Change from Baseline | SF-36 Acute Score has means at Day -1 and Day 7 | SAC[2] |
| Respir | atory Rate | | | | |
| 2.71 | All Subject | Non-Standard<br>EFF_F20 | Individual Plot of 24-Hour Respiratory Monitoring | There will be a graph for each patient individually | SAC[2] |
| 2.72 | All Subject | Non-Standard<br>EFF_F21 | Mean (95% CI) Plot of 24 Hour Respiratory Rate Monitoring | | SAC[2] |

# 11.13.7. Safety Tables

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Exposi | ure | | | | |
| 3.01 | All Subjects | EX1 | Summary of Extent of Exposure | | SAC [2] |
| Advers | se Events | | | | |
| 3.02 | All Subjects | AE5 | Summary of All Adverse Events by System Organ Class | Include total column. Exclude pre-treatment AEs and washout period AEs | SAC [2] |
| 3.03 | All Subjects | AE3 | Summary of Common Adverse Events by Overall Frequency | AE is considered common if more than one subject experiences it regardless of treatment. Exclude pre-treatment AEs and washout period AEs | SAC [2] |
| 3.04 | All Subjects | AE5 | Summary of Drug-Related Adverse Events by System Organ Class | Include total column. Exclude pre-treatment and washout period AEs | SAC [2] |
| 3.05 | All Subjects | AE1 | Summary of Serious Adverse Events by System Organ Class | | SAC [2] |
| 3.06 | All<br>Subjects | AE1 | Summary of Adverse Events Leading to Withdrawals from Study / Permanent Discontinuation of Study Treatment | | SAC [2] |
| 3.07 | All Subjects | AE15 | Summary of Common (>=20%) Non-serious Adverse<br>Events by System Organ Class and Preferred Term | | SAC [2] |
| 3.08 | All Subjects | AE16 | Summary of Serious Adverse Events by System<br>Organ Class and Preferred Term | | SAC [2] |

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labs | Labs | | | | |
| 3.09 | All Subjects | LB1 | Summary of Clinical Chemistry Laboratory Values by Visit | | SAC [2] |
| 3.10 | All Subjects | LB1 | Summary of Chemistry Changes from Baseline by Visit | | SAC [2] |
| 3.11 | All Subjects | LB3 | Summary of Chemistry Results by Potential Clinical Importance Criteria | | SAC [2] |
| 3.12 | All Subjects | LB2 | Summary of LFTs of Potential Clinical Importance by Visit | Include ALT and total Bilirubin | SAC [2] |
| 3.13 | All Subjects | LB1 | Summary of Percent Change from Baseline of LFTs by Visit | | SAC [2] |
| 3.14 | All Subjects | LB1 | Summary of Haematology/Coagulation Changes from Baseline by Visit | | SAC [2] |
| 3.15 | All Subjects | LB17 | Summary of Haematology Results by Potential Clinical Importance Criteria | | SAC [2] |
| Vital S | igns | | | | |
| 3.16 | All Subjects | VS1 | Summary of Vital Signs by Visit | Include the Respiration Rate and Temperature | SAC [2] |
| 3.17 | All Subjects | VS3 | Summary of Change from Baseline in Vital Signs by Visit | Include the Respiration Rate and Temperature | SAC [2] |
| 3.18 | All Subjects | VS2 | Summary of Vital Signs Results by Potential Clinical Importance Criteria | | SAC [2] |

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| ECGs | ECGs | | | | |
| 3.19 | All Subjects | EG1 | Summary of ECG Findings by Visit | | SAC [2] |
| 3.20 | All Subjects | EG2 | Summary of Maximum QTc Values by Category. | | SAC [2] |
| 3.21 | All Subjects | EG2 | Summary of Change from Baseline in ECG Values by Visit. | | SAC [2] |

#### 11.13.8. Pharmacokinetic Tables

| Pharma | Pharmacokinetic Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Co | ncentration Da | ta | | | |
| 4.01 | PK | PK01 | Summary of Plasma GSK2798745 Pharmacokinetic Concentration-Time Data (ng/mL) | | SAC [2] |
| 4.02 | Per<br>Protocol | PK01 | Summary of Plasma GSK2798745 Pharmacokinetic Concentration-Time Data (ng/mL) | Add Footnote | SAC [2] |
| PK Der | ived Paramete | ers | | | |
| 4.03 | 4.03 PK Parameter PKPT1 Summary Statistics of Derived Plasma GSK2798745 Pharmacokinetic Parameters Pharmacokinetic Parameters | | | | |
| 4.05 | PK<br>Parameter | PKPT3 | Summary Statistics of Log-Transformed Derived Plasma GSK2798745 Pharmacokinetic Parameters | Parameters with units | SAC [2] |

# 11.13.9. Pharmacokinetic Figures

| Pharma | Pharmacokinetic Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Individ | Individual Plots | | | | |
| 4.01 | PK | PKCF1P | Individual GSK2798745 Plasma Concentration-Time Plot by Treatment (Linear and Semi-Log) | Paginate by Treatment | SAC [2] |
| Mean / | Mean / Median Plots | | | | |
| 4.02 | PK | PKCF2 | Mean Plasma GSK2798745 Concentration-Time Plots by Treatment (Linear and Semi-log) | Paginate by Treatment | SAC [2] |

# 11.13.10. ICH Listings

| ICH Lis | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Rando | Randomisation | | | | |
| 01 | All Subjects | TA2 | Listing of Randomised and Actual Treatments | | SAC [2] |
| Subjec | t Disposition | | | | |
| 02 | All Subjects | ES3 | Listing of Reasons for Study Withdrawal | | SAC [2] |
| 03 | All Subjects | ES7 | Listing of Reasons for Screening Failure | | SAC [2] |
| 04 | All Subjects | SA3b | Listing of Subjects Excluded from Per Protocol Population | Only list subject that deviate from per protocol | SAC [2] |
| 05 | All Subjects | DV2 | Listing of Important Protocol Deviations | | SAC [2] |
| 06 | All Subjects | IE4 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC [2] |
| Demog | raphics | | | | |
| 07 | All Subjects | DM4 | Listing of Demographic Characteristics | | SAC [2] |
| 08 | All Subjects | DM10 | Listing of Race | | SAC [2] |
| Medica | Medical Conditions & Concomitant Medication | | | | |
| 09 | All Subjects | MH3 | Listing of Medical Conditions (Current/Past) | | SAC [2] |
| 10 | All Subjects | CM5 | Listing of Concomitant Medication | | SAC [2] |

| ICH Lis | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Exposi | Exposure | | | | |
| 11 | All Subjects | EX4 | Listing of Exposure | | SAC [2] |
| Advers | se Events | | | | |
| 12 | All Subjects | AE9 | Listing of All Adverse Events | | SAC [2] |
| 13 | All Subjects | AE9 | Listing of Serious Adverse Events | Only include AE's classified as serious | SAC [2] |
| 14 | All Subjects | AE9 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment. | | SAC [2] |
| 15 | All Subjects | ECSSRS4 | Listing of C-SSRS | | SAC [2] |
| 16 | All Subjects | EFF_L1 | Listing of SNAQ | | SAC [2] |
| 17 | All Subjects | EFF_L1 | Listing of Audiometry | | SAC [2] |
| 18 | All Subjects | EFF_L1 | Listing of Faecal Occult | | SAC [2] |
| Labs | | | | | |
| 19 | All Subjects | LB6 | Listing of Haematology Laboratory Data for Subjects with Abnormalities of Potential Clinical Importance | | SAC [2] |
| 20 | All Subjects | LB6 | Listing of Clinical Chemistry Laboratory Data for<br>Subjects Abnormalities of Potential Clinical<br>Importance | | SAC [2] |

| ICH Lis | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 21 | All Subjects | LB6 | Listing of LFT's for Subjects Abnormalities of Potential Clinical Importance | | SAC [2] |
| 22 | All Subjects | LB6 | Listing of Clinical Chemistry Laboratory Data for<br>Subjects Abnormalities of Potential Clinical<br>Importance As a Change from Baseline | Rather than have the value and normal range column just include a change from baseline column | SAC [2] |
| 23 | All<br>Subjects | LB6 | Listing of Haematology Laboratory Data for Subjects with Abnormalities of Potential Clinical Importance As a Change from Baseline | Rather than have the value and normal range column just include a change from baseline column | SAC [2] |
| ECGs | | | | | |
| 24 | All<br>Subjects | EG4 | Listing of ECG Values for Subjects with Abnormalities of Potential Clinical Importance. | | SAC [2] |
| Vital Si | gns | | | | |
| 25 | All<br>Subjects | VS5 | Listing of Vital Signs for Subjects with Abnormalities of Potential Clinical Importance | | SAC [2] |
| 26 | All<br>Subjects | VS5 | Listing of Vital Signs for Subjects | | SAC [2] |

# 11.13.11. Non-ICH Listings

| Non-IC | Non-ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Efficac | Efficacy | | | | |
| 28 | All Subjects | Non-Standard<br>EFF_L1 | Listing of Gas Diffusion Outcomes (DLco, DLno, Dm, Vc) | | SAC [2] |
| 29 | All Subjects | Non-Standard<br>EFF_L2 | Listing of Gas Diffusion Outcomes Change from Baseline (DLco, DLno, Dm, Vc) | | SAC [2] |
| 30 | All Subjects | Non-Standard<br>EFF_L1 | Listing of VE/VCO <sub>2</sub> | Rows for day -1 and day 7 only | SAC [2] |
| 31 | All Subjects | Non-Standard<br>EFF_L2 | Listing of VE/VCO <sub>2</sub> Change from Baseline | Rows for day -1 and day 7 only | SAC [2] |
| 32 | All Subjects | PFT9 | Listing of Pulmonary Function Test (FVC, FEV1, FEF-25-75, FEF50, FEF75) | Rows for day -1, day 4, and day 7 only | SAC [2] |
| 33 | All Subjects | Non-Standard<br>EFF_L2 | Listing of Pulmonary Function Test Change from Baseline (FVC, FEV1, FEF-25-75, FEF50, FEF75) | Rows for day -1, day 4, and day 7 only | SAC [2] |
| 34 | All Subjects | LB6 | Listing of Troponin | (Include change from baseline) | SAC [2] |
| 35 | All Subjects | SF6 | Listing of SF-36 Acute Score | | SAC [2] |
| 36 | All Subjects | MOS_S7 | Listing of Sleep Study Variables | Include Minimum Oxygen Saturation during sleep, total sleep time, central apnea index, obstructive apnea index, mixed apnea index, hypopnea index, apnea hypopnea index | SAC[2] |

| Non-ICH Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 40 | All Subjects | EFF_L2 | Listing of Change in Minimum Oxygen Saturation during Polysomnography | | SAC[2] |
| 41 | All Subjects | EFF_L1 | Listing of AUC of HMG-CoA reductase inhibitors and their key metabolites | | SAC[2] |
| 37 | All Subjects | SF6 | Listing of Dyspnea Score | (Include change from baseline) | SAC[2] |
| PK | | | | | |
| 38 | PK | PKCL1P | Listing of Plasma GSK2798745 Pharmacokinetic Concentration-Time Data | | SAC [2] |
| 39 | PK | PKPL1P | Listing of Derived Plasma GSK2798745 Pharmacokinetic Parameters | Include dose and dose number | SAC [2] |

# 11.14. Appendix 12: Example Mock Shells for Data Displays


Protocol : 201881 Population : All Subjects

Figure 1.1
Spaghetti Plot of DLco Data
DLco by Patient




Protocol : 201881 Population : All Subjects

Figure 1.02 Mean (95% CI) Plot of DLco

#### Mean DLCO per Visit, by Treatment




: EFF\_F3 Example Protocol : 201881 Population : All Subjects

Figure 1.03 Mean (95% CI) Plot of DLco

# Mean Chronic DLco by Treatment Group




Example : EFF\_F4
Protocol : 201881
Population : All Subjects

Figure 1.04 Plot of DLco by Individual and Treatment

#### DLco Over Time by Treatment Group




Example : EFF\_F5
Protocol : 201881
Population : All Subjects

Figure 1.05
Change from Baseline DLco by Individual and Treatment




Protocol : 201881
Population : All Subjects

Figure 1.06
Mean Plot of DLco Change from Baseline

# Mean Change from Baseline DLco by Treatment Group


Example : EFF\_F7
Protocol : 201881
Population : All Subjects

Figure 1.07
Mean Plot of DLco Pre/Post Exercise

## Mean DLco Pre/Post Exercise by Treatment Group



Example : EFF\_F8
Protocol : 201881
Population : All Subjects

Figure 1.08
Mean Plot of DLco Change from Exercise

## Mean Change from Exercise DLCO by Treatment Group



Example : EFF\_F9
Protocol : 201881
Population : All Subjects

Figure 1.09
Mean Plot of Percent Change DLco from Exercise

## Mean Percent Change from Exercise DLCO by Treatment Group



Example : EFF\_F10
Protocol : 201881
Population : All Subjects

Figure 1.10
Mean Plot of Percent Change DLco from Saline

## Mean Percent Change from Saline DLCO by Treatment Group




Protocol : 201881 Population : All Subjects

Figure 1.11 Plot of VE/VCO<sub>2</sub>

#### VE/VCO2 Ratio




Protocol : 201881 Population : All Subjects

Figure 1.12 Mean (95% CI) Plot of VE/VCO<sub>2</sub>

## Average Ve/VCO2 Ratio by Treatment




Protocol : 201881 Population : All Subjects

Figure 1.13 Plot of VE/VCO<sub>2</sub> Change from Day -1

## Change from Day -1 VE/VCO2 Ratio



Example : EFF\_F14
Protocol : 201881
Population : All Subjects

Figure 1.14
Plot of Mean VE/VCO<sub>2</sub> Change from Day -1

# Average Change from Day -1 Ve/VCO2 Ratio by Treatment



Example : EFF\_F15
Protocol : 201881
Population : All Subjects

Figure 1.15 Plot of VE/VCO<sub>2</sub> Change from Rest

### VE/VCO2 Ratio Change from Rest




Protocol : 201881 Population : All Subjects

Figure 1.16
Plot of Mean VE/VCO<sub>2</sub> Change from Rest

## Mean VE/VCO2 Ratio Change from Rest



Example : EFF\_F17
Protocol : 201881
Population : All Subjects

Figure 1.17 Spaghetti Plot of FVC



Example : EFF\_F18
Protocol : 201881
Population : All Subjects

Figure 1.18 Mean (95% CI) Plot of FVC



Example : EFF\_F19
Protocol : 201881
Population : All Subjects

Figure 1.19
Mean (95% CI) Plot of FVC Change from Baseline




Protocol : 201881 Population : All Subjects

Figure 1.20 Individual Plot of 24-Hour Respiratory Monitoring



Example : EFF\_F21
Protocol : 201881
Population : All Subjects

Figure 1.21
Mean (95% CI) Plot of 24 Hour Respiratory Rate Monitoring



Example : EFF\_F22
Protocol : 201881
Population : All Subjects

Figure 1.22 DLco Spaghetti Plot by Site





Example : EFF\_F23
Protocol : 201881
Population : All Subjects

Figure 1.23 Forest Plot of End Points



NOTE: Plot adjusted accordingly to study data, text values are the mean change from baseline.

Example : EFF\_F24
Protocol : 201881
Population : All Subjects

Figure 1.24 Dlco Saline Challenge Graph



NOTE: Plot adjusted accordingly to study data. The text is the difference between before and after and the percent change

Example : EFF\_T1
Protocol : 201881
Population : Analysis

#### Table 1.01 Summary Statistics of DLco

| Visit | Treatment | N | n | Mean | SD | Mean Percent<br>Predicted | Percent<br>Predicted SD |
|---|---|---|---|---|---|---|---|
| Screen | | Χ | Х | XX.X | XX.XX | XX.X | XX.XX |
| Baseline | Α | Х | Х | XX.X | XX.XX | | |
| Baseline after exercise | Α | Χ | Χ | XX.X | XX.XX | | |
| Day 4 | Α | Χ | Χ | XX.X | XX.XX | | |
| Day 5 | Α | Χ | Χ | XX.X | XX.XX | | |
| Day 5 after saline infusion | Α | Χ | Χ | XX.X | XX.XX | | |
| Day 7 | Α | Χ | Χ | XX.X | XX.XX | | |
| Day 7 after exercise | Α | Χ | Χ | XX.X | XX.XX | | |
| Baseline | В | Χ | Х | XX.X | XX.XX | | |
| Baseline after exercise | В | Χ | Χ | XX.X | XX.XX | | |
| Day 4 | В | Χ | Χ | XX.X | XX.XX | | |
| Day 5 | В | Χ | Χ | XX.X | XX.XX | | |
| Day 5 after saline infusion | В | Χ | Χ | XX.X | XX.XX | | |
| Day 7 | В | Χ | Χ | XX.X | XX.XX | | |
| Day 7 after exercise | В | Χ | Χ | XX.X | XX.XX | | |
| Follow-up | NA | Χ | Х | XX.X | XX.XX | | |

201881


Example : EFF\_T2
Protocol : 201881
Population : Analysis

Table 1.02 Summary Statistics of DLco Change from Baseline

| Visit | Treatment | N | n | Mean | SD |
|-----------------------------|-----------|---|---|------|-------|
| Baseline after exercise | Α | Х | X | XX.X | XX.XX |
| Day 4 | Α | Χ | Х | XX.X | XX.XX |
| Day 5 | Α | Χ | Χ | XX.X | XX.XX |
| Day 5 after saline infusion | Α | Χ | Χ | XX.X | XX.XX |
| Day 7 | Α | Χ | Χ | XX.X | XX.XX |
| Day 7 after exercise | А | X | Χ | XX.X | XX.XX |
| Baseline after exercise | В | Х | X | XX.X | XX.XX |
| Day 4 | В | Χ | Χ | XX.X | XX.XX |
| Day 5 | В | Χ | Χ | XX.X | XX.XX |
| Day 5 after saline infusion | В | Χ | Χ | XX.X | XX.XX |
| Day 7 | В | Χ | Χ | XX.X | XX.XX |
| Day 7 after exercise | В | Χ | Χ | XX.X | XX.XX |

201881


Example : EFF\_T3
Protocol : 201881
Population : Analysis

#### Table 1.03 Summary Statistics of DLno

| Visit | Treatment | N | n | Mean | SD |
|-----------------------------|-----------|---|---|------|-------|
| Screen | | Χ | Χ | XX.X | XX.XX |
| Baseline | Α | Χ | Х | XX.X | XX.XX |
| Baseline after exercise | Α | Χ | Χ | XX.X | XX.XX |
| Day 4 | Α | Χ | Χ | XX.X | XX.XX |
| Day 5 | Α | Χ | Χ | XX.X | XX.XX |
| Day 5 after saline infusion | Α | Χ | Χ | XX.X | XX.XX |
| Day 7 | Α | Χ | Χ | XX.X | XX.XX |
| Day 7 after exercise | Α | Χ | Χ | XX.X | XX.XX |
| Baseline | В | Χ | Χ | XX.X | XX.XX |
| Baseline after exercise | В | Χ | Χ | XX.X | XX.XX |
| Day 4 | В | Χ | Χ | XX.X | XX.XX |
| Day 5 | В | Χ | Χ | XX.X | XX.XX |
| Day 5 after saline infusion | В | Χ | Χ | XX.X | XX.XX |
| Day 7 | В | Χ | Χ | XX.X | XX.XX |
| Day 7 after exercise | В | Χ | X | XX.X | XX.XX |
| Follow-up | NA | Х | Х | XX.X | XX.XX |

201881

Example Protocol : EFF\_T4 : 201881 Page 1 of X

Population : Analysis

Table 1.04 Summary Statistics of FVC

| Visit | Treatment | N | n | Mean | SD |
|-----------|-----------|---|---|------|-------|
| Baseline | А | Χ | Χ | XX.X | XX.XX |
| Day 4 | Α | Χ | Χ | XX.X | XX.XX |
| Day 7 | Α | Χ | Χ | XX.X | XX.XX |
| Baseline | В | Х | Χ | XX.X | XX.XX |
| Day 4 | В | Χ | Χ | XX.X | XX.XX |
| Day 7 | В | Χ | Χ | XX.X | XX.XX |
| Follow-up | NA | Χ | Χ | XX.X | XX.XX |

201881

Example : EFF\_T5 Page 1 of X Protocol : 201881

Protocol : 201881
Population : Analysis

### Table 1.05 Summary Statistics of FVC Change from Baseline

| Visit | Treatment | N | n | Mean | SD |
|-------|-----------|---|---|------|-------|
| Day 4 | А | Χ | Χ | XX.X | XX.XX |
| Day 7 | Α | Χ | Χ | XX.X | XX.XX |
| Day 4 | В | X | Χ | XX.X | XX.XX |
| Day 7 | В | Χ | Χ | XX.X | XX.XX |

201881


Protocol : 201881 Population : Analysis

> Table 1.06 Summary of Statistical Analysis Results of DLco

Adjusted Mean

Treatment Placebo Difference Estimate 95% CI

XX.XX XX.XX XX.XX (XX.XX, XX.XX)

NOTE: Table adjusted accordingly to the study data, with model details added as footnotes.

201881


Example : EFF\_T7
Protocol : 201881

Population

: Analysis

Table 1.07 Summary Statistics of Ve/VCO2 Ratio

| Period | Sequence | Treatment | N | Visit | Mean At Rest | SD At Rest | Mean Post<br>1 Min | SD Post 1<br>Min | Mean Post<br>2 Min | SD Post 2<br>Min | Mean Post<br>3 Min | SD Post 3<br>Min | Mean<br>Recovery | SD<br>Recovery |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 1 | AB | Α | Х | Baseline | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX |
| | | Α | Χ | Day 7 | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX |
| 2 | AB | В | Χ | Baseline | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX |
| | | В | Χ | Day 7 | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX |
| Follow-up | AB | NA | Χ | Follow-up | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX |
| 1 | ВА | В | Χ | Baseline | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX |
| | | В | Χ | Day 7 | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX |
| 2 | BA | Α | Χ | Baseline | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX |
| | | Α | Χ | Day 7 | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX |
| Follow-up | BA | NA | Χ | Follow-up | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX |

201881


Example Protocol : EFF\_T8 : 201881

Population : Analysis

### Table 1.08 Summary Statistics of Ve/VCO2 Ratio Change from Baseline

| Period | Sequence | Treatment | N | Visit | Mean At<br>Rest | SD At<br>Rest | Mean Post<br>1 Min | SD Post 1<br>Min | Mean Post<br>2 Min | SD Post 2<br>Min | Mean Post<br>3 Min | SD Post 3<br>Min | Mean<br>Recovery | SD<br>Recovery |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 1 | AB | Α | Χ | Day 7 | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX |
| 2 | AB | В | Χ | Day 7 | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX |
| Follow-up | AB | NA | Χ | Follow-up | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX |
| 1 | ВА | В | Χ | Day 7 | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX |
| 2 | ВА | Α | Χ | Day 7 | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX |
| Follow-up | BA | NA | Χ | Follow-up | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X | XX.XX |

201881

Example : EFF\_T9 : 201881 Page 1 of X

Protocol Population : Analysis

#### Table 1.09 Summary Statistics of Dyspnea

| Visit | Treatment | N | n | Mean | SD | Median | Range | Percent of Patients with at Least 1- Point Improvement <sup>1</sup> | I | Frequen | cy of Itei | m Score: | s |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | 1 | 2 | 3 | 4 | 5 |
| Baseline Pre-Exercise | Α | Χ | Χ | XX.X | XX.XX | XX.X | X - X | | Χ | Χ | Χ | Χ | Χ |
| Baseline Post-Exercise | Α | Χ | Χ | XX.X | XX.XX | XX.X | X - X | XX.XX | Χ | Χ | Χ | Χ | Χ |
| Day 5 Sitting | Α | Χ | Χ | XX.X | XX.XX | XX.X | X - X | XX.XX | Χ | Χ | Χ | Χ | Χ |
| Day 5 Supine | Α | Χ | Χ | XX.X | XX.XX | XX.X | X - X | XX.XX | Χ | Χ | Χ | Χ | Χ |
| Day 7 Pre-Exercise | Α | Χ | Χ | XX.X | XX.XX | XX.X | X - X | XX.XX | Χ | Χ | Χ | Χ | Χ |
| Day 7 Post-Exercise | Α | Χ | Χ | XX.X | XX.XX | XX.X | X - X | XX.XX | Χ | Χ | Χ | Χ | Χ |
| Baseline Pre-Exercise | В | Χ | Χ | XX.X | XX.XX | XX.X | X - X | | Χ | Χ | Χ | Χ | Χ |
| Baseline Post-Exercise | В | Χ | Χ | XX.X | XX.XX | XX.X | X - X | XX.XX | Χ | Χ | Χ | Χ | Χ |
| Day 5 Sitting | В | Χ | Χ | XX.X | XX.XX | XX.X | X - X | XX.XX | Χ | Χ | Χ | Χ | Χ |
| Day 5 Supine | В | Χ | Χ | XX.X | XX.XX | XX.X | X - X | XX.XX | Χ | Χ | Χ | Χ | Χ |
| Day 7 Pre-Exercise | В | Χ | Χ | XX.X | XX.XX | XX.X | X - X | XX.XX | Χ | Χ | Χ | Χ | Χ |
| Day 7 Post-Exercise | В | Χ | Χ | XX.X | XX.XX | XX.X | X - X | XX.XX | Χ | Χ | Χ | Χ | Χ |
| Follow-up | NA | Χ | Χ | XX.X | XX.XX | XX.X | X - X | | Χ | Χ | Χ | Χ | Χ |

201881


Protocol : 201881 Population : Analysis

Table 1.11

Summary Statistics of Respiratory Rate

Day -1 Day 4 Day 7

Placebo Placebo Treatment Placebo Treatment Treatment Mean SD Number of Mean SD Number of SD Number of Mean SD Number of SD Number of SD Number of Mean Mean Mean Hours Hours Hours Hours Hours Hours Included Included Included Included Included Included

Lying Standing Leaning

201881


Example : EFF\_T12
Protocol : 201881
Population : Analysis

Table 1.12 Summary Statistics of DLco Change from Intervention

| Visit | Treatment | N | n | Mean | SD |
|-----------------------------------|-----------|---|---|------|-------|
| Baseline change from exercise | Α | Χ | Χ | XX.X | XX.XX |
| Day 5 change from saline infusion | Α | Χ | Χ | XX.X | XX.XX |
| Day 7 change from exercise | Α | Χ | Χ | XX.X | XX.XX |
| Baseline change from exercise | В | Х | X | XX.X | XX.XX |
| Day 5 change from saline infusion | В | Χ | Χ | XX.X | XX.XX |
| Day 7 change from exercise | В | Χ | Χ | XX.X | XX.XX |

201881

Example : EFF\_L1 Page 1 of X Protocol : 201881

Population : All Subjects

Listing 1 Listing of Gas Diffusion

| Sequence | Treatment | Subject | Visit | DLco | DLno | $D_M$ | VE/VCO <sub>2</sub> |
|---|---|---|---|---|---|---|---|
| AB | | 1 | Screening | | | | |
| | | | Period 1 Baseline | | | | |
| | Α | | Period 1 Day -1 Post Exercise | | | | |
| | Α | | Period 1 Day 4 | | | | |
| | Α | | Period 1 Day 5 | | | | |
| | В | | Period 1 Day 5 Post-Saline | | | | |
| | | | Period 2 Baseline | | | | |
| | В | | Period 2 Day -1 Post Exercise | | | | |
| | В | | Period 2 Day 4 | | | | |
| | В | | Period 2 Day 5 | | | | |
| | В | | Period 2 Day 5 Post-Saline | | | | |

Follow-Up

201881

Example Protocol : EFF\_L2 Page 1 of X

Population : Safety

## Listing 2 Listing of Gas Diffusion Change from Baseline

| Sequence | Treatment | Subject | Visit | Change<br>in DLco | Change<br>in DLno | Change<br>in D <sub>M</sub> | Change<br>in<br>VE/VCO <sub>2</sub> |
|---|---|---|---|---|---|---|---|
| AB | A<br>A<br>A | | Period 1 Day -1 Post Exercise Period 1 Day 4 Period 1 Day 5 Period 1 Day 5 Post-Saline | | | | |
| | B<br>B<br>B | | Period 2 Day -1 Post Exercise<br>Period 2 Day 4<br>Period 2 Day 5<br>Period 2 Day 5 Post-Saline | | | | |